## Protocol A6181213

# **RENACALL**

Evaluation of the impact of a call center in management of metastatic and/or advanced renal cell carcinoma patients treated with sunitinib (Sutent) in first line

Prospective, multicenter usual care study conducted in mainland France

## Statistical analytical plan (SAP)

| Sponsor: Pfiz | er |
|-----------------|---------------------|
| Medical lead | s: PPD |
| Project leads | : PPD |
| CRO: PPD | |
| Scientific Dire | ector: Dr PPD |
| Project leads | :PPD |
| Biostatisticia | n/Data Manager: PPD |
| Version: | Final version (FV) |
| Author: | PPD |
| Date: | 06 February 2019 |

| Scientific Committee Coordinator: |
|-----------------------------------|
| Dr PPD |
| Medical Oncologist |
| PPD |
| Scientific Committee: |
| Dr PPD |
| Medical Oncologist |
| PPD |
| Dr PPD |
| Medical oncologist |
| PPD |
| Prof. PPD |
| Professor in Public Health |
| PPD |

## **TABLE OF CONTENTS**

| 1. | VERS | SION HISTORY | 9 |
|---|---|---|---|
| 2. | INTR | RODUCTION | 10 |
| 2. | .1. | Justification for the study | 10 |
| 2. | .2. | Plan of the study | 10 |
| 2. | .3. | Objectives | 13 |
| 3. | INTE | RIM ANALYSIS AND FINAL ANALYSIS | 14 |
| 4. | НҮР | OTHESES AND DECISION-MAKING RULES | 15 |
| 4. | .1. | Hypotheses | 15 |
| 4. | .2. | Decision-making rules | 15 |
| 5. | ANA | LYSIS POPULATION | 16 |
| 5. | .1. | Definition of the analysis populations | 16 |
| 5. | .2. | Analysis subgroup | 17 |
| 6. | END | POINTS | 18 |
| 6. | .1. | Primary end point | 18 |
| 6. | .2. | Secondary end points | 18 |
| 7. | MAN | NAGEMENT OF MISSING VALUES | 19 |
| 8. | STAT | FISTICAL METHODOLOGY AND STATISTICAL ANALYSES | 20 |
| 8. | .1. | Statistical methods | 20 |
| 8. | .2. | Statistical analyses | 21 |
| 9. | RESU | JLTS | 33 |
| 9. | .1. | Numbers | 33 |
| 9. | .2. | Description of the population when sunitinib treatment is started | 39 |
| 9. | .3. | Description of patients during the follow-up period | 49 |
| 9. | .4. | Analysis of the primary end point | 57 |
| 9. | .5. | Analysis of the secondary end points | 58 |
| 9. | .6. | Pharmacovigilance | 74 |
| 9. | .7. | Supplementary analysis: Patient follow-up "Standard follow-up" | 77 |
| 10. | RE | EFERENCES | 82 |
| 11. | Ar | nnexes | 83 |

| 11.1. | Interpretation of the Kappa coefficient | 83 |
|---|---|---|
| 11.2. | Definition of region indicators | 84 |
| list of t | ables | |
| List of t | ables | |
| Table 1: F | Patient eligibility criteria | 11 |
| Table 2: [ | Data collected during the RENACALL study inclusion and follow-up consultations | 12 |
| Table 3: F | Population in each analysis | 16 |
| Table 4: ( | Characteristics of participating and non-participating investigators | 33 |
| Table 5: 0 | Characteristics of active investigators | 34 |
| Table 6: F | Reasons for non-inclusion of patients entered into the non-inclusion register | 35 |
| Table 7: 0 | Characteristics of included and non-included patients | 36 |
| Table 8: [ | Description of patient follow-up | 36 |
| | nclusion characteristics of patients who were followed up and those who were not follow | |
| Table 10: | Sociodemographic characteristics of patients (safety population) at inclusion | 39 |
| Table 11: | Clinical characteristics of patients (safety population) at inclusion | 39 |
| Table 12: | Description of the patients' primary renal cell carcinoma (safety population) at inclusion. | 40 |
| | Description of the treatment of the patients' primary renal cell carcinoma (safety on) at inclusion | 40 |
| | Description of the patients' advanced/metastatic renal cell carcinoma (safety population | |
| | Past medical history and previous or current comorbidities of patients (safety population | |
| Table 16: | Treatments being received at inclusion for ongoing comorbidities (safety population) | 42 |
| Table 17: | Hematologic profile before starting the Sunitinib (safety population) | 43 |
| Table 18: | Biochemical profile before starting Sunitinib (safety population) | 44 |
| | Abnormal values for other hematologic and biochemical indices before starting Sunitinib | |
| Table 20: | Other patient investigations (safety population) at inclusion | 47 |

| Table 21: Symptomatic or preventative treatments prescribed (safety population) at inclusion 48 |
|---|
| Table 22: Supportive measures for sunitinib treatment (safety population) at initiation 48 |
| Table 23: Description of changes to treatment with sunitinib in terms of dosage and dosage regimen (safety population - Call Center |
| Table 24: Tumor assessments (safety population - Call Center) during the follow-up period 49 |
| Table 25: Clinical indices (safety population - Call Center) during the follow-up period |
| Table 26: Hematologic and biochemical profile (safety population - Call Center) during the follow-up period |
| Table 27: Abnormal values for other hematologic and biochemical indices (safety population - Call Center) during the follow-up period |
| Table 28: Symptoms of patients who were followed up (safety population - Call Center) during the follow-up period |
| Table 29: Supportive measures for sunitinib treatment (safety population - call center follow-up) during the follow-up period, instituted by the doctor |
| Table 30: Development of AEs during the follow-up period (safety population) |
| Table 31: Description of grade 3 and 4 AEs related or unrelated to sunitinib recorded during the follow-up period (safety population) |
| Table 32: Description of dose reductions (safety population) |
| Table 33: Dose reductions made depending on the number of calls received (safety population) 58 |
| Table 34: Description of temporary interruption of sunitinib treatment during the follow-up period (safety population) |
| Table 35: Temporary interruption of sunitinib treatment during the follow-up period depending on number of calls received (safety population) |
| Table 36: Description of discontinuations of sunitinib treatment during the follow-up period (safety population) |
| Table 37: Requirements for medical procedures by cycle during the follow-up period (safety population) |
| Table 38: Number of medical procedures per cycle during the follow-up period (safety population) 61 |
| Table 39: Morisky scale items during the follow-up period (safety population) |
| Table 40: Assessment of adherence during the follow-up period (safety population) |
| Table 41: Morisky scale items in week 4 of cycles 1, 2 and 4 (safety population)64 |

| Table 42: Assessment of adherence in week 4 of cycles 1, 2 and 4 (safety population) 64 |
|---|
| Table 43: Consistency between assessment of adherence at W4 (telephone) and W6 (self-completed questionnaire) in each cycle 1, 2 and 4 (safety population) |
| Table 44: Response to sunitinib treatment (FAS population) |
| Table 45: Frequency of calls made during sunitinib treatment by cycle and overall (FAS population) 67 |
| Table 46: Actions by doctors and patients assessed during the first call (FAS population) |
| Table 47: Actions by doctors and patients assessed during the first call in cycles 2, 3 and 4 (FAS population) |
| Table 48: Advice given during calls by the support call center by cycle and overall (FAS population). 68 |
| Table 49: Satisfaction of doctors who included patients followed up by the call center with the patient treatment management call center |
| Table 50: Characteristics of doctors who were satisfied or very satisfied with the support from the patient treatment management call center |
| Table 51: Satisfaction of patients included in the Call Center arm with the call center (FAS Call Center population) |
| Table 52: Other satisfaction indicators for patients included in the Call Center arm with the call center (FAS Call Center population) |
| Table 53: Caracteristics of patients who were satisfied or very satisfied with the support, in patients in the Call Center arm (FAS Call Center population) |
| Table 54: Description of all of the AEs declared during the study (Safety population) |
| Table 55: Description of all AEs related to sunitinib declared during the follow-up period (Safety population) |
| Table 56: Tumor assessments (safety population- standard follow-up) during the follow-up period . 77 |
| Table 57: Clinical indices (safety population- standard follow-up) during the follow-up period 77 |
| Table 58: Symptoms (safety population- standard follow-up) during the follow-up period |
| Table 59: Supportive measures for sunitinib treatment (safety population- standard follow-up) during the follow-up period, instituted by the doctor |
| Table 60: Follow-up data(safety population- standard follow-up) |
| Table 61: Requirement for medical procedures (safety population- standard follow-up) |
| Table 62: Patient adherence with treatment (safety population- standard follow-up) |

# List of figures

| Figure 1: Plan of telephone calls | 10 |
|----------------------------------------------------------|----|
| Figure 2: Numbers of investigators | 33 |
| Figure 3: Flow-chart of patient numbers during the study | 35 |
| Figure 4: Definition of region indicators | 84 |

## **Abbreviations**

| a/mRCC | Advanced/metastatic renal cell carcinoma |
|---------|------------------------------------------------|
| AEs | Adverse Events |
| ALT | Alanine Transaminase |
| ANOVA | Analysis of variance |
| AST | Aspartate Transaminase |
| ВМІ | Body Mass Index |
| CATI | Computer-assisted telephone interview |
| СС | follow-up by a "call center" |
| CI | Confidence Interval |
| CRO | Clinical Research Organization |
| CTCAE | Common Terminology Criteria for Adverse Events |
| ECG | Electrocardiogram |
| ECO CRU | Health Economics Clinical Research Unit |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic Case Report Form |
| GEE | Generalized Estimating Equations |
| нт | Hypertension |
| INCA | French National Cancer Institute |
| INFα | Alpha interferon |
| ITT | Intention to Treat |
| IV | Intravenous |
| MAR | Missing At Random |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMAS | Morisky Medication Adherence Scale |
| NB | Negative Binomial |
| ORR | Objective Response Rate |
| PT | Preferred Term |
| PV | Pharmacovigilance |
| QC | Quality Control |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SD | Standard Deviation |
| SF | Standard follow-up |
| SmPC | Summary or product characteristics |
| SOC | System Organ Class |
| SOP | Standard Operating Procedures |
| ZIP | Zero-Inflated Poisson |
| ZNB | Zero-inflated Negative Binomial |

## 1. VERSION HISTORY

| Version | Amendments | Date |
|---------|---------------|------------|
| V6.3 | Final version | 06/02/2019 |

## 2. INTRODUCTION

The introduction to this document briefly summarizes the main features of the RENACALL study on the basis of the amendment to the protocol No. 3.1 of 21 July 2017. Items shown in italics originate from this protocol.

To recall, this last amended version removes of the concept of randomization into two follow-up arms and discontinues the "standard follow-up" arm.

## 2.1. Justification for the study

Cell therapy treatment requires close patient monitoring to ensure the medicinal product is used correctly, and particularly to prevent and manage adverse events (AEs). Improved management of adverse events helps to optimize the duration of treatment and the clinical benefit of treatment. Most of the targeted therapies are taken orally and the adverse events often occur at home. Regular contact by a treatment management call center could not only reduce the percentage of patients developing a grade 3-4 adverse event but also reduce the number of unplanned hospitalizations and consultations due to poor tolerability.

No studies have assessed the impact of follow-up using a "treatment management call center" on the treatment of patients suffering from metastatic/advanced renal cell carcinomas treated with a targeted oral therapy. Improvement in the care of patients treated with an oral targeted therapy is one of the priorities in the  $2^{nd}$  cancer plan produced by INCa (http://www.plan-cancer.gouv.fr/).

The RENACALL study is designed to assess a method for managing patients under real life conditions which is different from usual follow-up, with no additional interventions of the part of the doctor.

## 2.2. Plan of the study

## General plan

The RENACALL study is a prospective, multicenter, usual care study conducted in Mainland France in adult patients suffering from advanced/metastatic renal cell carcinoma treated first line with sunitinib. The study will be conducted in 10 to 20 centers which look after renal cancer.

The therapeutic management of patients within the facility will not be changed by the study and will follow the recommendations in the SmPC. Patients who are included will receive an additional intervention with follow-up from the treatment management telephone call center. Management through the treatment management telephone call center involves regular telephone calls (cf. Figure 1) in order to support the patient in his/her home management with sunitinib treatment under real life conditions (prevention, advice and directing patients towards options available).



Figure 1. Plan of telephone calls

## Populations

## Population of Participating doctors

The study will be proposed to 58 doctors throughout 50 Mainland France oncology centers identified as treating patients suffering from metastatic/advanced renal cell carcinoma. It is planned to identify 20 to 25 doctors liable to take part in the study.

These centers will be selected by the Pfizer Company. They will need to have a number of patients which meet the eligibility criterion which is sufficient to be included (approximately 10 patients per year) and not to have a routine management call center already in place in their facility.

#### Patient Population

**Inclusion criteria** 

It is expected to recruit 100 patients for this study, i.e. approximately 10 per center. The patients must meet the following inclusion and non-inclusion criteria.

Non-inclusion criteria

Table 1: Patient eligibility criteria

#### - Men or women, aged 18 years old or over; - Patients taking part in a clinical trial during - Patients suffering from advanced and/or treatment with sunitinib; - Patients managed by a home hospitalization service metastatic renal cell carcinoma treated first line with sunitinib according to the SmPC during treatment with sunitinib; recommendations; - Patients taking part in therapeutic education - Starting Sutent® in accordance with the SmPC programs or receiving a nurse consultation or any recommendations (50 mg/day, dosage regimen other significant support for treatment liable to 4/2); impact on the management of adverse effects; - Resolution (grade ≤ 1 according to CTCAE version Patients suffering from untreated and/or 4.03 dated June 2010) of all the acute toxic effects symptomatic cerebral metastases before beginning due to previous treatment with radiotherapy or a sunitinib: - Patients who refuse to allow their personal data to surgical procedure before starting sunitinib; - Patients who can be followed up for 6 months; be used: - Patients of childbearing potential who must be - Patients with an ECOG performance index at using a method of contraception throughout the inclusion > 2; period of treatment with sunitinib and for a - Patients with a serum creatinine of > 1.5 times the minimum of 28 days after stopping treatment with upper limit of normal; - Patients with bilirubin concentrations > 2 mg/dl, - Patients who have given their signed consent; aspartate transaminase (AST) or alanine transaminase (ALT) levels > 2.5 times the upper limit of normal - Patients belonging to a social security system. value or > 5 times the upper limit of normal in the presence of liver metastases when sunitinib treatment is started; - Patients who are staff members of the center involved in the study or are personal friends to a member of the center directly involved in the management of the study, or patients who are employed by Pfizer and are involved in the conduct of the study.

## Data collection

The data collected during the inclusion and follow-up visits are shown in Table 2:

Table 2: Data collected during the RENACALL study inclusion and follow-up consultations

| | V0: Inclusion T0 | V1: end of<br>cycle 1<br>W6 | V2: end of<br>cycle 2<br>W12 | V3: end of<br>cycle 4<br><i>W24</i> |
|---|---|---|---|---|
| Data completed by the doctor (in the eCRF) | | | | |
| Meeting the eligibility criteria | х | | | |
| ECOG performance index | х | х | Х | х |
| Karnofsky index/Heng criterion risk score | х | | | |
| Sociodemographic features | х | | | |
| History of the disorder/description of the renal cell | х | | | |
| carcinoma | | | | |
| Past medical history and comorbidities | х | | | |
| Tumor assessment/ Disease assessment | | х | х | х |
| Data from the laboratory, histological or metastatic | х | х | х | х |
| assessments | | | | |
| Conditions for the use of Sunitinib | х | | | |
| Change in the conditions of use for Sunitinib | | х | Х | х |
| Concomitant treatments | х | х | Х | х |
| Pharmacovigilance data | | х | Х | х |
| Medical procedures (telephone calls, consultations, | | х | Х | х |
| hospitalizations), both planned and unplanned | | | | |
| Issuing of support materials for treatment with sunitinib | х | х | х | х |
| Data completed by the patient (self-completed questi | ionnaire) | | | |
| Adherence to treatment (4 item Morisky | | х | х | х |
| questionnaire) | | | | |
| Data completed by the doctor (in the eCRF) and patier | nt (self-completed | questionnaire) | | |
| Satisfaction with the telephone call center | | | | Х |

The following data will be collected by the nurses during the telephone calls (recorded by a CATI - Computer-Assisted Telephone Interview) system:

- Number of attempts and outcome of the call;
- General patient health;
- Administration of treatment;
- Tolerability and onset of AEs (description of the AE: intensity, symptoms, impact on the patient, investigations, action instituted);
- Proposed action.

The investigator characteristics will be obtained from an extraction from the database provided by Pfizer.

## 2.3. Objectives

## **Primary objective**

- To assess the impact of a treatment management call center on the treatment of patients suffering from advanced/metastatic renal cell carcinoma (a/mRCC) treated 1<sup>st</sup> line with sunitinib.

## Secondary objectives

- To describe and estimate the proportion of patients who have dose reductions, interruptions or discontinuation of treatment (Sutent®),
- To estimate the number of unplanned medical procedures, whether or not related to Sutent® (number of unplanned consultations and hospitalizations),
- To assess adherence with treatment (Morisky scale [1, 2]),
- To estimate the objective response rate (ORR) according to RECIST criteria v1.1.
- To assess patient and doctor satisfaction with the telephone call center,
- To describe the process of the telephone calls in terms of the number of calls completed and actions taken by the call center and/or the doctor.

## 3. INTERIM ANALYSIS AND FINAL ANALYSIS

No interim analysis is planned.

The **final data analysis** will be performed following the data collection and after freezing the database as approved with Pfizer. After the amendment to the protocol (no. 3.1), it was agreed that the statistical analyses be performed on all patients who were followed up by the telephone "Call Center" platform.

Patients initially included in the "standard follow-up" group will be described for informative purposes from their major characteristics at inclusion and during follow-up.

A final statistical report will describe all of the planned analyses in the SAP and any additional analyses requested. This statistical report will not contain any description or comment about the results.

A study report will be written and submitted to Pfizer. This document will provide a discussed overview of the results of the analyses in order to meet the objectives of the study.

The results of the RENACALL study may be discussed in terms of the results of the SANTORIN study [8].

The reports will be written in French.

## 4. HYPOTHESES AND DECISION-MAKING RULES

## 4.1. Hypotheses

No statistical tests will be used.

## 4.2. Decision-making rules

Not applicable.

## 5. ANALYSIS POPULATION

## **5.1.** Definition of the analysis populations

Reported population 
All patients reported by the investigators in the non-inclusion register and

included in the eCRF.

**Safety population** Patients treated with Sunitinib.

Full Analysis Set (FAS)

All patients included by the investigating doctors who meet the study

**Population** eligibility criteria and have received at least one dose of Sunitinib

**NB:** Where applicable, the two subgroups of patients will in all cases be distinguished in the populations: firstly patients included in the "Call Center" arm (main interest population) and patients included in the "standard follow-up" arm (exploratory population) set up as part of the initial study design (before amendment No. 3 to the protocol).

Table 3: Population in each analysis

| Analyses | | Populations analyzed | Analysis subgroup* |
|---|---|---|---|
| Description at inclusion | | Safety population | Call Center /standard follow-up |
| Description of follow-up | All data | Safety population Call Center | |
| | Main data | Safety population Standard follow-up | |
| Primary objective | | Safety population | Number of calls made by the call center* |
| Secondary objectives | Sunitinib treatment details | Safety population | Number of calls made by the call center* |
| | Planned and unplanned medical procedures | Safety population | Number of calls made by the call center* |
| | Adherence to treatment | Safety population | Number of calls made by the call center* |
| | Objective response rate | FAS population | Number of calls made by the call center* |
| | Telephone calls | Call Center FAS population | |
| | Patient satisfaction | Call Center FAS population who completed a self-administered satisfaction questionnaire | Number of calls made by the call center* |
| | Doctor satisfaction | Call Center FAS population for which the<br>Doctors have completed a satisfaction<br>questionnaire | |
| Pharmacovigilance | | Safety population | |

<sup>\*</sup> cf. definition §5.2.

## 5.2. Analysis subgroup

In the assessment of the treatment call center for patient management, analysis of the objectives may be performed overall and according to the number of calls received (two group classification).

In order to define compliance or non-compliance with the intervention, i.e. in order to define the patient as having actually followed the procedure, the scientific committee will define a minimum number of 7 successful calls out of the planned 14 calls over 4 cycles, with a required minimum of 6 successful calls during the first two treatment cycles, representing at least 3 calls in each of the first two cycles.

## 6. END POINTS

## 6.1. Primary end point

The primary end point is defined as the percentage of patients with at least one grade 3 or 4 adverse event (whether or not related to Sutent®), during the first 4 cycles of treatment (study follow-up period) according to the 'Common Terminology Criteria for Adverse Events' (CTCAE) version 4.03 of June 2010).

## 6.2. Secondary end points

## - Dose reductions, interruptions and discontinuations of treatment (sunitinib)

#### **Description of dose reductions:**

- Proportion of patients with at least one dose reduction compared to the initial dose:
- Reasons for dose reductions;
- Changes in dose (initial dose or new prescribed dose).

## **Description of treatment interruptions:**

- Proportion of patients who temporarily interrupt sunitinib;
- Mean duration of interruptions;
- Reasons for interruptions.

#### Permanent discontinuation of treatment

- Proportion of patients who discontinue Sunitinib permanently;
- Reasons for discontinuations.

## Unplanned medical procedures:

- Average number of unplanned consultations, whether or not related to sunitinib;
- Average number of unplanned hospitalizations, whether or not related to sunitinib.

#### Treatment adherence

Adherence to treatment will be assessed from the **mean adherence score** and from the **proportion of "adherent" patients.** These criteria will be determined using the **Morisky scale** (**MMAS-4**: 4-item Morisky Medication Adherence Scale), which consists of 4 items, together with a further question about adverse effects completed by the patient.

#### Response to treatment

Response to treatment will be assessed from the **objective response rate (ORR)** according to RECIST criteria V1.1.

#### Patient and doctor satisfaction with the telephone call center

Patient satisfaction with the call center will be assessed by:

- the mean scores for each dimension on the satisfaction questionnaire;
- the proportion of patients/doctors who reported being "satisfied" or "very satisfied" overall with the management by the telephone call center.

## - Description of telephone calls

The telephone calls received during the study will be described by:

- the number of completed calls (planned and unplanned),
- the actions taken by the patient,
- the actions taken by the call center,
- the actions taken by the doctor,
- and the declaration of adverse events.

## 7. MANAGEMENT OF MISSING VALUES

The data from patients were recorded on an eCRF, except for the paper self-completed adherence and patient satisfaction questionnaires. Mandatory fields and consistency controls will be used to check data registered at the time. This strategy will be used to reduce missing data points or inconsistencies, particularly those concerning the major end points (AE, grades of AE and response to treatment etc.).

The analyses will be performed on the available data ("observed case analysis"), using the assumption that missing data are non-informative. The numbers of missing data points will be presented for each variable.

The response analysis will also be conducted on the FAS population by imputing missing responses as failure (= progression).

## 8. STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

The statistical analyses will be performed on SAS software (version 9.4 or subsequent, SAS Institute, North Carolina USA).

#### 8.1. Statistical methods

## 8.1.1. Descriptive analyses

The analysis will be purely descriptive.

The descriptive analysis of qualitative variables will include numbers and frequency of each modality. The analysis of quantitative variables will include mean, standard deviation, values, median and extreme values. The number of missing values or values analyzed will be shown for each variable studied.

Consistency between two qualitative variables (assessment of adherence at W4 and W6 of cycles 1, 2 and 4) will be assessed using the Kappa coefficient [3] (cf. interpretation of the Kappa coefficient in annex 11.1).

## 8.1.2. Analysis strategy

In the principal analysis of the primary objective, all patients included in the "Call Center" arm will be analyzed in this group regardless of the number of calls received and all of their data will be used.

The analysis will be performed on an overall basis and according to the number of calls made by the call center as defined in section §5. Analysis population.

The statistical analyses and tabular models stipulated in this SAP will be used subject to sufficient numbers being available for the expanded analysis for a given variable.

## 8.2. Statistical analyses

#### 8.2.1. **Numbers**

The numbers of participating investigating doctors will be described, together with the average number of patients included in the study. Participating and non-participating investigators will be described by geographical region (a variable derived from the post code of the investigator: cf. annex 1). The characteristics of active and non-active investigators will be described by geographical region, type of practice, urban or non-urban area and age and sex. The type of center facility will also be described (general hospital, university hospital, cancer center, etc.). These data will be obtained from an extraction from the database provided by Pfizer.

The **patient numbers** during the study will be displayed in a flow chart (cf. Figure 3 on page 35): patients reported, patients included, those followed up, those which leave the study and those who die.

Eligible patients who are not included into the study will be described from the data collected in the non-inclusion register in parallel with the same characteristics as patients who are included: age (derived from date of birth), sex and ECOG performance index. The reasons for non-inclusion will also be presented.

Follow-up of patients who are included will be described by:

- The median follow-up time in weeks: the time between the date of the inclusion visit and the date of the last follow-up consultation (If a patient stops treatment permanently during the follow-up period after the patient has stopped treatment will be included for patients in the CC arm).
- Average number of treatment cycles per patient;
- Average number of follow-up consultations achieved per patient;
- Average number completed calls per patient in the CC arm.

The major inclusion characteristics of patients who were followed up and those who were not followed up will be presented.

# 8.2.2. Description of the population when sunitinib treatment is started

**Population analyzed:** Included population

## **Analysis:**

The patients will be described when they start treatment with sunitinib from all of the **inclusion data** collected:

- Patients' sociodemographic characteristics: Age (calculated as the time in years between date of birth and date of starting sunitinib), and sex;
- Clinical Characteristics of the patients: Risk score Heng et al. criteria, Body Mass Index (BMI), ECOG performance index and Karnofsky index;
- History of the disorder: Time since the initial diagnosis of the primary renal cell carcinoma (calculated as the time in years between the date of initial diagnosis and the date of starting sunitinib), histology, stage of the disease, Fuhrman grade, treatment for the primary renal cell carcinoma (nephrectomy, radiotherapy or other), time since diagnosis of the 1<sup>st</sup> metastases (calculated as the time in years between the date of diagnosis of the 1<sup>st</sup> metastases and the date of starting sunitinib) and site of the metastases;
- Past medical history: Previous or ongoing comorbidities (diabetes, thyroid, etc.);
- Hematologic and biochemical profile before starting sunitinib: Time since the laboratory profile (in days), values of indices assessed (hemoglobin, platelets, LDH, etc.), abnormal values for other indices (hematocrit, leucocytes, etc.);
- Other investigations performed: Blood pressure, electrocardiogram (ECG), echocardiogram and previous orodental examination;
- Concomitant symptomatic or preventative treatments: Antiemetic or anti-diarrheal treatment, anti-neutropenic treatment, etc.;
- Treatment supportive measures: Person delivering the information on treatment, issuing of materials/support or document to the patient.

## 8.2.3. Description of patients during the follow-up period

## **Populations analyzed:**

- Safety population: Call Center (all data) and standard follow-up (main data)

## **Analysis:**

On an exploratory basis, before the analysis of the study objectives, the patients will be described from the data completed during the follow-up period by the investigating doctor:

- Tumor assessment: Radiologic investigation, response to treatment;
- Clinical parameters: ECOG, Karnofsky index and blood pressure;
- Hematologic and biochemical profile: Values of the indices measured (hemoglobin, calcium, etc.) and abnormal values for other indices (hematocrit, leucocytes, etc.);
- Symptoms and tolerability: Development of AEs: gastrointestinal or cardiac problems, etc.; Description serious AEs and non-serious AEs.
- Concomitant, symptomatic or preventative treatments: Prescription of another additional anti-tumor treatment, antiemetic treatment, anti-diarrheal treatment, etc.;
- Planned and unplanned medical procedures: number of calls, consultations and hospitalizations performed, specialty of the health professional in the event of calls or consultations, duration of hospitalization, reason for the medical procedure (AE or other) and actions implemented;
- Measures to support treatment when treatment is continued: Person delivering the information about treatment, issuing of materials/supports or documents to the patient.

The data listed above will be described for each follow-up time (end of cycle 1, 2 and 4).

## 8.2.4. Analysis of the primary end point

**Analysis population**: Safety population

The proportion of patients with at least one grade 3 or 4 AE whether or not related to sunitinib, will be estimated.

All of the grades 3 or 4 AEs defined by the 'Common Terminology Criteria for Adverse Events' (CTCAE v4.03 of June 2010), whether or not related to sunitinib, will be included when these occur during the study follow-up period (up to the end of the 4<sup>th</sup> treatment cycle or until the treatment is stopped if it is discontinued in the 1<sup>st</sup>, 2<sup>nd</sup> or 3<sup>rd</sup> cycle). All of the AEs will be included whether these are declared by the doctor or by the nurse.

The analyses will be performed both on an overall basis and according to the number of calls made by the call center.

#### **Sensitivity analyses:**

The sensitivity analyses will be performed:

• Sensitivity to duration of patient treatment: the results will also be expressed as standardized grade 3 or 4 AE rates developed by the patient and reported over the 6 months of treatment. These rates will be defined by each patient as the number of events which occurred/number of treatment months with sunitinib/ 6).

## **Secondary analysis:**

The incidence of the main grade 3 or 4 AEs, whether or not related to sunitinib, will also be
presented in these patients according to the MedDRA SOC (System Organ Class) and PT
(Preferred Term) classification. Only categories involving at least 2% of patients will be
presented.

## 8.2.5. Analysis of the secondary end points

#### 8.2.5.1. Sunitinib treatment

**Populations analyzed:** Safety population

#### **End points:**

The analysis of sunitinib treatment methods will be carried out using the following indicators:

#### Description of dose reductions

- Proportion of patients with at least one dose reduction during the period of sunitinib treatment:
- Reasons for the dose reduction: Proportion of patients involved on at least one occasion for each of the reasons for a dose reduction;
- Average dose reduction.

#### Description of interruptions to treatment

- Proportion of patients who interrupted sunitinib treatment temporarily during treatment (including declared temporary interruptions and cases in which the start of the later cycle was deferred);
- Mean duration (in days) of interruptions to treatment by patient (declared duration of interruption or number of days delay identified for the start of the subsequent cycle);
- Reason for interruptions: Proportion of patients involved on at least one occasion for each of the reasons for interruption of treatment (AE, radiotherapy, surgery or other).

## Description of permanent treatment discontinuations

- Proportion of patients who discontinued sunitinib permanently;
- Reason for discontinuation: proportion of patients involved on at least one occasion for each of the reasons for discontinuation;
- Duration of treatment with sunitinib: time between starting sunitinib and the notified date to discontinue it or the date of the last consultation if sunitinib treatment was not stopped;
- o Number of treatment cycles before discontinuation.

The analysis will be performed both on an overall basis and according to the number of calls made by the call center.

# 8.2.5.2. Number of unplanned medical procedures, whether or not related to Sunitinib

Analysis population: Safety population

## **Analysis:**

The purpose of estimating the number of unplanned medical procedures particularly involves those unplanned consultations and hospitalizations, whether or not related to sunitinib and declared at each follow-up visit.

At each theoretical follow-up time (end of cycles 1, 2 and 4 and overall), the following indicators will be described on an overall basis:

- Proportion with at least 1 consultation, at least 1 hospitalization, resulting in at least 1 planned or unplanned call to a health professional;
- Average number of consultations and hospitalizations (two different indicators) both planned and unplanned and the total number per cycle per patient;
- Total number of consultations and hospitalizations (single indicator) by cycle during sunitinib treatment. The number of planned, unplanned and the total number of calls to a health professional by cycle, by patient will also be described for descriptive purposes.

The analysis will be performed on an overall basis and by the number of calls made by the call center.

## 8.2.5.3. Adherence to treatment

**Population analyzed:** Safety population

#### **Analysis:**

Adherence to sunitinib treatment will be assessed from the standardized, validated, Morisky self-completed questionnaire (MMAS-4: 4-item Morisky Medication Adherence Scale), completed by the patients at the 6 wee follow-up visit in cycles 1, 2 and 4. This questionnaire consists of 4 items each with two response options "Yes" and "No".

An **MMAS-4 score** will be calculated as the number of "Yes" responses and will be between 0 and 4, a low score representing improved adherence. The score will be missing if one of the items has not been completed.

A classification using the MMAS-4 score will be used to categorize adherence into levels [3; 4]:

- High adherence: score of 0;
- Average adherence: score of 1 or 2;
- Poor adherence: score of 3 or 4.

At each measurement time (end of cycles 1, 2 and 4), the following indicators will be described:

- average adherence score;
- proportion of patients by a patient adherence level;
- the proportion of "adherent" patients, defined as patients with an MMAS score of 0 and the proportion of "non-adherent" patients as patients with a score of at least 1 [6].
- An assessment of patient behavior in terms of their treatment when they develop an AE (binary indicator (Yes/No) for reduction or adjustment of treatment).

In order to examine the change in adherence by patient, the mean difference in patient score between the assessment at the end of cycle 1 and the assessment at cycle 4 will be described.

The analysis will be performed on an overall basis and by the number of calls made by the call center.

<u>In addition and only for informative purposes</u>, the Morisky questionnaire will also be completed through the call center during the call on W4 of cycles 1, 2 and 4 and in the "Call Center" group. This assessment will be used:

- firstly to measure adherence at the end of the 4<sup>th</sup> week of treatment (immediately before the treatment break) from the derived criteria described above (average score, proportion of adherent patients);
- secondly, to estimate (subject to sufficient numbers being available) good consistency between patient declarations between the measurement on W4 and the consultation on W6 during which the patient will complete his/her self-administered questionnaire.

Concordance will only be measured for informative purposes as the questionnaire has been validated for self-completion by the patient him/herself and not as one administered by a third party (potential declaration bias concerning the issue of adherence).

The MMAS-4 score ranges from 0 to 4 (discrete quantitative variable), and can be considered to be qualitative index. Consistency between adherence at week 4 assessed by telephone and adherence at week 6 assessed in writing will be considered using the Kappa coefficient.

## 8.2.5.4. Response to sunitinib treatment

**Analysis population:** FAS population

## **Analysis:**

The response to treatment will be assessed by the investigator based on RECIST v1.1 criteria (complete response, partial response, stable disease or progression) and will be described at each follow-up time (at the end of cycles 1, 2 and 4) (cf. section 8.2.3. Description of patients during the follow-up period).

The best response obtained during treatment with sunitinib will be identified from the responses assessed according to RECIST v1.1 criteria. "Unevaluable" responses will not be included in the definition of the best response.

The proportion of patients with a complete or partial best response during the follow-up period (objective response rate) will be estimated.

The last response assessed during the study will also be estimated.

The analysis will be performed on an overall basis and by the number of calls made by the call center.

Analysis of response will also be assessed on the FAS population imputing missing data points by failure (= progression).

## 8.2.5.5. Telephone calls made

## **Analysis population:**

- FAS population, regardless of the number of calls completed.
- All calls made.

## **Analysis:**

The average number of planned, unplanned and the total number of calls made per patient will be presented on an overall basis and by treatment cycle.

The conduct of the telephone calls will be described using the following indicators:

- Action taken by the patient;
- And/or action taken by the doctor;
- Declaration of adverse events;
- o Action taken by the call center.

#### 8.2.5.6. Doctor satisfaction with the call center

<u>Analysis population:</u> FAS population for which the Doctors have completed a satisfaction questionnaire

#### **Analysis:**

The doctor's satisfaction with the call center will be assessed from the doctor satisfaction questionnaire which will be completed by the doctors at the end of the follow-up period.

This questionnaire, which has been constructed for the study, is made up of 5 questions with responses in the form of a semantic odd number measurement scale (5 modalities: "Very unsatisfied", "satisfied", "not particularly satisfied", "unsatisfied" and "no opinion"), including 3 satisfaction dimensions (overall satisfaction, satisfaction with the advice given and satisfaction with the management).

Each response is allocated a positive or negative score (+2, +1, -1, -2 and no score) respectively allowing a quantitative score to be established for each item. A score will be calculated for each dimension of the questionnaire by calculating the mean scores obtained for each item if at least 50% of the items for the dimension have been completed (and are not "no opinion").

The doctor's satisfaction with the call center will be assessed from:

- The mean score for each dimension: A radar plot with 3 axes will be proposed in order to simultaneously show the mean scores for each dimension. In this type of display, the mean scores are linked together and form a polygon. The area of the polygon will be described and the ratio between the area of the polygon and the ratio of the ideal polygon (complete coverage of the radar plot) will be used to assess the percentage surface area covered. A high area represents better general satisfaction.
- The proportion of doctors who reported themselves as being "Very satisfied" or "Satisfied" overall with management by the call center (5<sup>th</sup> item of the questionnaire).

These doctors will be described by sex, age and number of patients in the CC arm before being involved with the call center when at least 50% of the planned calls are completed.

#### 8.2.5.7. Patient satisfaction with the call center

<u>Analysis population:</u> FAS population included in the Call Center arm who completed a self-administered satisfaction questionnaire.

#### **Analysis:**

The patient satisfaction analysis with the call center will be assessed from the self-administered satisfaction questionnaire completed at the end of the study by each patient in the CC arm. This questionnaire together with the doctor questionnaire has been created for this study.

The questionnaire contains 8 items, and is theoretically completed during the final visit at week 6 of cycle 4. For patients who stop their treatment at the end of cycles 1, 2 or 3, the questionnaire will be completed in the last follow-up visit performed (the visit in which discontinuation of treatment is notified).

Definition of scores by dimension (overall satisfaction with advice, satisfaction with the service and satisfaction with the management) will be similar to what is described in the previous section "doctor satisfaction with the call center".

Patient satisfaction with the call center will be assessed from:

- The mean scores for each dimension; a radar plot with 4 axes will be proposed in order to simultaneously represent the mean scores for each dimension. In the same manner as for the assessment of doctor's satisfaction, the area of the polygon and percentage of subjects covered will be described.
- The proportion of patients who reported themselves as being "Very satisfied" or "Satisfied" overall with the support offered by the call center (8<sup>th</sup> item of the questionnaire).

These patients will be described by their major characteristics when they started sunitinib (sex, age, ECOG score, etc.).

## 8.2.6. Pharmacovigilance

**Analysis population:** Safety population

#### Analysis:

The proportion of patients who develop at least one adverse event whether or not related to Sunitinib will be described.

All of the adverse events declared during the study will be described from:

- Their title (coded according to MedDRA);
- The time (in days) between starting sunitinib and the onset of the AE;
- The severity of the adverse effect;
- Its grade;
- Impact on everyday activities;
- Causality;
- Corrective medical action;
- Last actions taken for sunitinib during the AE.

Before the database is frozen, the listing of AEs and SAEs will be provided to the Pfizer Company, in order to undertake a reconciliation between the Kappa Santé and the Pfizer data.

The pharmacovigilance indicators described above will be provided for each of the following AE groups:

- All of the AEs (regardless of severity);
- Non-serious AEs;
- Serious AEs.

#### 8.2.7. Listings

Patient listings will be provided in the annex to the statistical report when specific cases exist such as the following situations:

- Patients excluded from the analysis (Patient no. + reason for exclusion);
- Patients with AEs and SAEs;
- Patients with dosage reductions, changes, interruptions or discontinuation.

## 9. RESULTS

## 9.1. Numbers

## 9.1.1. Investigators



Figure 2: Numbers of investigators

The active centers included an average of xx patients into the study (min: xx; max: xx).

Table 4: Characteristics of participating and non-participating investigators

| | | Participating investigators | |
|---|---|---|---|
| | | Yes | No |
| | | (N=xxx) | (N=xxx) |
| Geographical region* | PPD | xx (xx%) | xx (xx%) |
| | | xx (xx%) | xx (xx%) |
| Facility | General Hospital | xx (xx%) | xx (xx%) |
| • | University Hospital | xx (xx%) | xx (xx%) |
| | Private Clinic | xx (xx%) | xx (xx%) |
| | Cancer Center | xx (xx%) | xx (xx%) |
| | Other | xx (xx%) | xx (xx%) |
| | Not stated | xx - | xx - |

<sup>\*</sup> Derived from the center post code (cf. annex 1)

**Table 5: Characteristics of active investigators** 

| | | Active inve | estigators |
|----------------------|---------------------|-------------|------------|
| | | Yes | No |
| | | (N=xxx) | (N=xxx) |
| Geographical region* | PPD | xx (xx%) | xx (xx%) |
| | | xx (xx%) | xx (xx%) |
| Facility | General Hospital | xx (xx%) | xx (xx%) |
| | University Hospital | xx (xx%) | xx (xx%) |
| | Private Clinic | xx (xx%) | xx (xx%) |
| | Cancer Center | xx (xx%) | xx (xx%) |
| | Other | xx (xx%) | xx (xx%) |
| | Not stated | xx - | xx - |
| Type of practice | Primary Care | xx (xx%) | xx (xx%) |
| | Hospital | xx (xx%) | xx (xx%) |
| | Mixed | xx (xx%) | xx (xx%) |
| | Not stated | xx - | xx - |
| Urban environment | Yes | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) |
| | Not stated | xx - | xx - |
| Sex | Male | xx (xx%) | xx (xx%) |
| | Female | xx (xx%) | xx (xx%) |
| | Not stated | XX - | XX - |
| Age (years) | Number analyzed | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) |
| | Median | XX | XX |
| | Min-Max | xx - xx | xx - xx |

<sup>\*</sup> Derived from the center post code (cf. annex 1)

## 9.1.2. Patients



<sup>\*</sup>Non-inclusion register

Figure 3: Flow-chart of patient numbers during the study

Table 6: Reasons for non-inclusion of patients entered into the non-inclusion register

| | Patient refusal | Non-included patients<br>(N=xxx) |
|---|---|---|
| Reason for non-inclusion | | xx (xx%) |
| | Other | xx (xx%) |
| | Details | xx (xx%) |

Table 7: Characteristics of included and non-included patients

| | | Patients included | |
|---|---|---|---|
| | | Yes | No |
| | | (N=xxx) | (N=xxx) |
| Characteristics at inclusion | | | |
| Age (years) | Number<br>analyzed | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) |
| | Median | xx | xx |
| | Q1-Q3 | xx - xx | xx - xx |
| | Min-Max | xx - xx | xx - xx |
| Sex | Male | xx (xx%) | xx (xx%) |
| | Female | xx (xx%) | xx (xx%) |
| ECOG score | 0 | xx (xx%) | xx (xx%) |
| | 1 | xx (xx%) | xx (xx%) |
| | 2 | xx (xx%) | xx (xx%) |
| | 3 | xx (xx%) | xx (xx%) |
| | 4 | xx (xx%) | xx (xx%) |
| | Not stated | xx (xx%) | xx (xx%) |

Table 8: Description of patient follow-up

| | | Standard<br>follow-up<br>(N=xxx) | Call Center<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| | | | , | |
| Follow-up time (weeks) (time between inclusion and date | Number analyzed | xxx | xxx | xxx |
| of last follow-up consultation) | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| · | Median | xx | xx | xx |
| | Q1-Q3 | xx - xx | xx - xx | xx - xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Number of treatment cycles per patient | Number analyzed | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Mean duration of cycles 1 (days) | Number analyzed | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Mean duration of cycles 2 (days) | Number analyzed | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Mean duration of cycles 3 (days) | Number analyzed | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Mean duration of cycles 4 (days) | Number analyzed | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Number of follow-up consultations carried out per patient | Number analyzed | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Number of calls | Number analyzed | - | xxx | - |
| | Mean (±SD) | - | xx (± xx) | - |
| | Standard<br>follow-up<br>(N=xxx) | Call Center<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Median | - | xx | - |
| Min-Max | - | xx - xx | - |

Table 9: Inclusion characteristics of patients who were followed up and those who were not followed up

| | | Follow | ed up | Total |
|---|---|---|---|---|
| | | Yes | No | (N=xxx) |
| | | (N=xxx) | (N=xxx) | |
| haracteristics at inclusion | | | | |
| Age (years) | Number | xxx | xxx | xxx |
| | analyzed | | | |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Sex | Male | xx (xx%) | xx (xx%) | xx (xx%) |
| | Female | xx (xx%) | xx (xx%) | xx (xx%) |
| ECOG score | 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| | 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| | 2 | xx (xx%) | xx (xx%) | xx (xx%) |
| | 3 | xx (xx%) | xx (xx%) | xx (xx%) |
| | 4 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not stated | xx - | xx - | xx - |
| Risk score – Heng criteria | Good | xx (xx%) | xx (xx%) | xx (xx%) |
| · · | Intermediary | xx (xx%) | xx (xx%) | xx (xx%) |
| | Poor | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not available | xx (xx%) | xx (xx%) | xx (xx%) |
| Fuhrman grade | I | xx (xx%) | xx (xx%) | xx (xx%) |
| • | II | xx (xx%) | xx (xx%) | xx (xx%) |
| | III | xx (xx%) | xx (xx%) | xx (xx%) |
| | IV | xx (xx%) | xx (xx%) | xx (xx%) |
| Metastatic renal cell carcinoma grade | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Previous or current comorbidities | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |

## 9.2. Description of the population when sunitinib treatment is started

## 9.2.1. Sociodemographic characteristics

Table 10: Sociodemographic characteristics of patients (safety population) at inclusion

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Age (years) | Number analyzed | xxx | XXX | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | xx |
| | Q1-Q3 | xx - xx | xx - xx | xx - xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Sex | Male | xx (xx%) | xx (xx%) | xx (xx%) |
| | Female | xx (xx%) | xx (xx%) | xx (xx%) |

#### 9.2.2. Clinical Characteristics

Table 11: Clinical characteristics of patients (safety population) at inclusion

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Body Mass Index (BMI) | Lean: < 18,5 | xx (xx%) | xx (xx%) | xx (xx%) |
| , | Normal body weight: [18,5; 25[ | xx (xx%) | xx (xx%) | xx (xx%) |
| | Overweight: [25; 30[ | xx (xx%) | xx (xx%) | xx (xx%) |
| | Obese: ≥ 30 | xx (xx%) | xx (xx%) | xx (xx%) |
| ECOG score | 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| | 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| | 2 | xx (xx%) | xx (xx%) | xx (xx%) |
| | 3 | xx (xx%) | xx (xx%) | xx (xx%) |
| | 4 | xx (xx%) | xx (xx%) | xx (xx%) |
| Karnofsky index scored | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| · | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, Karnofsky index | 100% | xx (xx%) | xx (xx%) | xx (xx%) |
| | 90% - 80% | xx (xx%) | xx (xx%) | xx (xx%) |
| | 70% - 60% | xx (xx%) | xx (xx%) | xx (xx%) |
| | 50% - 40% | xx (xx%) | xx (xx%) | xx (xx%) |
| | 30% - 10% | xx (xx%) | xx (xx%) | xx (xx%) |
| | 0% | xx (xx%) | xx (xx%) | xx (xx%) |
| Risk score – Heng et al. criteria | Good | xx (xx%) | xx (xx%) | xx (xx%) |
| _ | Intermediary | xx (xx%) | xx (xx%) | xx (xx%) |
| | Poor | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not available | xx (xx%) | xx (xx%) | xx (xx%) |

#### 9.2.3. History of the disorder

Table 12: Description of the patients' primary renal cell carcinoma (safety population) at inclusion

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Time since initial diagnosis of the | Number analyzed | xxx | xxx | xxx |
| primary renal cell carcinoma | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| (years) | Median | XX | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Histology | Clear cell carcinoma | xx (xx%) | xx (xx%) | xx (xx%) |
| | Tubulo-papillary carcinoma | xx (xx%) | xx (xx%) | xx (xx%) |
| | Type I | xx (xx%) | xx (xx%) | xx (xx%) |
| | Type II | xx (xx%) | xx (xx%) | xx (xx%) |
| | Chromophobe cell carcinoma | xx (xx%) | xx (xx%) | xx (xx%) |
| | Other | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details | xx (xx%) | xx (xx%) | xx (xx%) |
| Mixed tumor | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, predominant tumor | Details | xx (xx%) | xx (xx%) | xx (xx%) |
| | ••• | xx (xx%) | xx (xx%) | xx (xx%) |
| Status of disease – TNM | TO | xx (xx%) | xx (xx%) | xx (xx%) |
| Classification | T1 | xx (xx%) | xx (xx%) | xx (xx%) |
| | T2 | xx (xx%) | xx (xx%) | xx (xx%) |
| | T3 | xx (xx%) | xx (xx%) | xx (xx%) |
| | T4 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Tx | xx (xx%) | xx (xx%) | xx (xx%) |
| | ND | xx (xx%) | xx (xx%) | xx (xx%) |
| | NO | xx (xx%) | xx (xx%) | xx (xx%) |
| | N1 | xx (xx%) | xx (xx%) | xx (xx%) |
| | N2 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Nx | xx (xx%) | xx (xx%) | xx (xx%) |
| | ND | xx (xx%) | xx (xx%) | xx (xx%) |
| | M0 | xx (xx%) | xx (xx%) | xx (xx%) |
| | M1 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Mx | xx (xx%) | xx (xx%) | xx (xx%) |
| | ND | xx (xx%) | xx (xx%) | xx (xx%) |
| Fuhrman grade | I | xx (xx%) | xx (xx%) | xx (xx%) |
| | II | xx (xx%) | xx (xx%) | xx (xx%) |
| | III | xx (xx%) | xx (xx%) | xx (xx%) |
| | IV | xx (xx%) | xx (xx%) | xx (xx%) |

Table 13: Description of the treatment of the patients' primary renal cell carcinoma (safety population) at inclusion

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Nephrectomy | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Radiotherapy | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Other treatment for cancer | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If other, treatment | Details | xx (xx%) | xx (xx%) | xx (xx%) |
| | | xx (xx%) | xx (xx%) | xx (xx%) |

Table 14: Description of the patients' advanced/metastatic renal cell carcinoma (safety population) at inclusion

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| etastatic renal cell carcinoma | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| ade | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes | | | | |
| Time since development of 1st | Number analyzed | XXX | XXX | XX |
| metastases (years) | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx |
| | Median | XX | XX | X |
| | Min-Max | xx - xx | xx - xx | xx - x |
| Number of different metastatic | Number analyzed | xx (xx%) | xx (xx%) | xx (xx% |
| sites involved | Mean (±SD) | xx (xx%) | xx (xx%) | xx (xx% |
| | Median | xx (xx%) | xx (xx%) | xx (xx% |
| | Min-Max | xx (xx%) | xx (xx%) | xx (xx% |
| Site of metastases | Lung | xx (xx%) | xx (xx%) | xx (xx% |
| | Bone | xx (xx%) | xx (xx%) | xx (xx% |
| | Mediastinum | xx (xx%) | xx (xx%) | xx (xx% |
| | Liver | xx (xx%) | xx (xx%) | xx (xx% |
| | Retroperitoneal lymph nodes | xx (xx%) | xx (xx%) | xx (xx% |
| | Supra-clavicular lymph nodes | xx (xx%) | xx (xx%) | xx (xx% |
| | Adrenal | xx (xx%) | xx (xx%) | xx (xx% |
| | Nephrectomy cavity | xx (xx%) | xx (xx%) | xx (xx% |
| | Kidney | xx (xx%) | xx (xx%) | xx (xx% |
| | Brain | xx (xx%) | xx (xx%) | xx (xx% |
| | Skin | xx (xx%) | xx (xx%) | xx (xx% |
| | Peritoneum | xx (xx%) | xx (xx%) | xx (xx% |
| | Gastro-intestinal | xx (xx%) | xx (xx%) | xx (xx% |
| | Pancreas | xx (xx%) | xx (xx%) | xx (xx% |
| | Other | xx (xx%) | xx (xx%) | xx (xx% |
| | Details | xx (xx%) | xx (xx%) | xx (xx% |
| If brain metastases, | Yes | xx (xx%) | xx (xx%) | xx (xx% |
| tumor untreated and/or symptomatic | No | xx (xx%) | xx (xx%) | xx (xx% |

# 9.2.4. Past medical history and comorbidities

Table 15: Past medical history and previous or current comorbidities of patients (safety population) at inclusion

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Comorbidities either previously | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| or at the time of inclusion | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, type | Diabetes | xx (xx%) | xx (xx%) | xx (xx%) |
| (several options possible) | Thyroid | xx (xx%) | xx (xx%) | xx (xx%) |
| | Hypothyroidism | xx (xx%) | xx (xx%) | xx (xx%) |
| | Hyperthyroidism | xx (xx%) | xx (xx%) | xx (xx%) |
| | CVA | xx (xx%) | xx (xx%) | xx (xx%) |
| | Hypertension | xx (xx%) | xx (xx%) | xx (xx%) |
| | Myocardial infarction | xx (xx%) | xx (xx%) | xx (xx%) |
| | Deep venous thrombosis | xx (xx%) | xx (xx%) | xx (xx%) |
| | Angina pectoris | xx (xx%) | xx (xx%) | xx (xx%) |
| | Renal impairment | xx (xx%) | xx (xx%) | xx (xx%) |
| | Hepatic impairment | xx (xx%) | xx (xx%) | xx (xx%) |
| | Other | xx (xx%) | xx (xx%) | xx (xx%) |
| Comorbidities ongoing at the | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| time inclusion | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, type | Diabetes | xx (xx%) | xx (xx%) | xx (xx%) |
| (several options possible) | Thyroid | xx (xx%) | xx (xx%) | xx (xx%) |
| | Hypothyroidism | xx (xx%) | xx (xx%) | xx (xx%) |
| | Hyperthyroidism | xx (xx%) | xx (xx%) | xx (xx%) |
| | CVA | xx (xx%) | xx (xx%) | xx (xx%) |
| | Hypertension | xx (xx%) | xx (xx%) | xx (xx%) |
| | Myocardial infarction | xx (xx%) | xx (xx%) | xx (xx%) |
| | Deep venous thrombosis | xx (xx%) | xx (xx%) | xx (xx%) |
| | Angina pectoris | xx (xx%) | xx (xx%) | xx (xx%) |
| | Renal impairment | xx (xx%) | xx (xx%) | xx (xx%) |
| | Hepatic impairment | xx (xx%) | xx (xx%) | xx (xx%) |
| | Other | xx (xx%) | xx (xx%) | xx (xx%) |

Table 16: Treatments being received at inclusion for ongoing comorbidities (safety population)

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Ongoing treatments (several options possible) | For: | | | |
| .,, | Diabetes | xx (xx%) | xx (xx%) | xx (xx% |
| | Thyroid | xx (xx%) | xx (xx%) | xx (xx% |
| | Hypothyroidism | xx (xx%) | xx (xx%) | xx (xx% |
| | Hyperthyroidism | xx (xx%) | xx (xx%) | xx (xx% |
| | CVA | xx (xx%) | xx (xx%) | xx (xx% |
| | Hypertension | xx (xx%) | xx (xx%) | xx (xx |
| | Myocardial infarction | xx (xx%) | xx (xx%) | xx (xx |
| | Deep venous thrombosis | xx (xx%) | xx (xx%) | xx (xx |
| | Angina pectoris | xx (xx%) | xx (xx%) | xx (xx |
| | Renal impairment | xx (xx%) | xx (xx%) | xx (xx |
| | Hepatic impairment | xx (xx%) | xx (xx%) | xx (xx |
| | Other | xx (xx%) | xx (xx%) | xx (xx |

## 9.2.5. Hematologic and biochemical profile

Table 17: Hematologic profile before starting the Sunitinib (safety population)

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Length of history (in months) from | Number analyzed | xxx | xxx | xxx |
| the last laboratory assessment | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| • | Median | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Hematologic profile | | | | |
| Hemoglobin | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | |
| Value (g/dL) | Number analyzed | XXX | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Neutrophils | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | |
| Value (mm³) | Number analyzed | XXX | XXX | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Platelets | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | |
| Value (10 <sup>9</sup> /L) | Number analyzed | XXX | XXX | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |

Table 18: Biochemical profile before starting Sunitinib (safety population)

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Length of history (in months) from | Number analyzed | xx (xx%) | xx (xx%) | xx (xx% |
| the last laboratory assessment | Mean (±SD) | xx (xx%) | xx (xx%) | xx (xx% |
| the last laboratory assessment | Median | <b>,</b> , | ( -/ | |
| | Min-Max | | | |
| Biochemical profile | | | | |
| Creatinine, (mg/dL) | Number analyzed | xxx | xxx | XX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx |
| | Median | XX | XX | X |
| | Min-Max | xx - xx | xx - xx | xx - x |
| ALT (SGPT) (U/L) | Number analyzed | xxx | xxx | xx |
| ALI (SGPI) (U/L) | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx |
| | Median | XX | XX | х |
| | Min-Max | xx - xx | xx - xx | xx - x |
| AST (SGOT) (U/L) | Number analyzed | XXX | XXX | XX |
| | Mean (±SD) | xx (± xx)<br>xx | xx (± xx)<br>xx | xx (± xx<br>x |
| | Median<br>Min-Max | xx - xx | xx - xx | xx - x |
| Bilirubin (mg/dL) | Number analyzed | XXX | XXX | XX |
| 5 (IIIg/ a.z/ | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx |
| | Median | XX | XX | × |
| | Min-Max | xx - xx | xx - xx | xx - x |
| Calcium | Value obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx% |
| If value obtained, | | xxx | xxx | xx |
| Value (mmol/L) | Number analyzed | | | |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx |
| | Median<br>Min-Max | xx<br>xx - xx | xx<br>xx - xx | xx - x |
| Albumin | Value obtained | xx (xx%) | xx (xx%) | xx (xx% |
| Albanini | Value not obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx% |
| If value obtained, | | | | |
| Value (g/L) | Number analyzed | XXX | XXX | XX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx |
| | Median | XX | XX | х |
| | Min-Max | xx - xx | xx - xx | xx - x |
| LDH | Value obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx% |
| If value obtained, | Number and | xxx | xxx | xx |
| Value (IU/L) | Number analyzed | xx (± xx) | xx (± xx) | xx (± xx |
| | Mean (±SD) | XX (± XX) | XX (± XX) | XX (I XX |
| | Median | | | |
| | Min-Max | xx - xx | xx - xx | xx - x |

Table 19: Abnormal values for other hematologic and biochemical indices before starting Sunitinib (safety population)

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Abnormal values for biological | Yes | xx (xx%) | xx (xx%) | xx (xx% |
| indices | No | xx (xx%) | xx (xx%) | xx (xx% |
| If yes, | | | | |
| Hematologic profile | | | | |
| Hematocrit | Value obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Value not obtained<br>Not performed | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) | xx (xx%<br>xx (xx% |
| If value obtained, | | | | |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx% |
| | No | xx (xx%) | xx (xx%) | xx (xx% |
| If result abnormal, | | | | |
| Value (%) | Number analyzed | XXX | XXX | XX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx |
| | Median | XX | XX | X |
| | Min-Max | xx - xx | xx - xx | XX - X |
| eucocytes | Value obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx% |
| If value obtained, | v | xx (xx%) | xx (xx%) | xx (xx% |
| abnormal result | Yes<br>No | xx (xx%) | xx (xx%) | xx (xx% |
| | INO | XX (XXX) | XX (XXX) | XX (XXX |
| If result abnormal, | | | | |
| Value (10 <sup>9</sup> /L) | Number analyzed | xxx<br>xx (± xx) | xxx<br>xx (± xx) | xx<br>xx (± xx |
| | Mean (±SD)<br>Median | XX (± XX) | XX (± XX) | XX (± XX |
| | Min-Max | xx - xx | xx - xx | xx - x |
| Biochemical profile | | | | |
| Alkaline phosphatase | Value obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx% |
| If value obtained, | | vv. (vv%) | vv (vv%) | vv (vv% |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx% |
| | No | xx (xx%) | xx (xx%) | xx (xx% |
| If result abnormal, | | | | |
| Value (U/L) | Number analyzed | xxx<br>xx (± xx) | XXX | xx (± xx |
| | Mean (±SD)<br>Median | XX (± XX) | xx (± xx)<br>xx | XX (± XX |
| | Min-Max | xx - xx | xx - xx | xx - x |
| TSH | Value obtained | xx (xx%) | xx (xx%) | xx (xx% |
| 1311 | Value not obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx% |
| If value obtained, | | | | |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx% |
| | No | xx (xx%) | xx (xx%) | xx (xx% |
| If result abnormal, | | | | |
| Value (mU/L) | Number analyzed | xxx | xxx | XX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx |
| | Median | XX | xx | X |
| | Min-Max | xx - xx | xx - xx | xx - x |
| fT3 | Value obtained | xx (xx%) | xx (xx%) | xx (xx% |

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx% |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If result abnormal, | | | | |
| Value (pmol/L) | Number analyzed | XXX | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | XX - XX |
| fT4 | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | / 0/> | / 0/> | ( 0() |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If result abnormal, | | | | |
| Value (pmol/L) | Number analyzed | XXX | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | XX - XX |
| Sodium | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | xx (xx%) | vv (vv%) | vv. (vv%) |
| abnormal result | Yes | ` ′ | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If result abnormal, | | | | |
| Value (mmol/L) | Number analyzed | XXX | xxx | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | XX - XX |
| Potassium | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | (9/) | /9/\ | /9/ |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If result abnormal, | | | | |
| Value (mmol/L) | Number analyzed | XXX | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | XX - XX | XX - XX |

## 9.2.6. Other investigations

Table 20: Other patient investigations (safety population) at inclusion

| | | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Blood pressure | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| • | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, | | xxx | xxx | xxx |
| Systolic value (mmHg) | Number analyzed | | | |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Diastolic value (mmHg) | Number analyzed | xxx | xxx | xxx |
| , , | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Electrocardiogram (ECG) | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| <u>If yes,</u> | | | | |
| Result normal | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| <u>If abnormal,</u> | Atrial fibrillation (AF) | xx (xx%) | xx (xx%) | xx (xx%) |
| (several responses are | Ventricular dysrhythmias | xx (xx%) | xx (xx%) | xx (xx%) |
| (several responses are<br>possible) | Atrio-ventricular block (AVB) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Other | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details<br> | xx (xx%) | xx (xx%) | xx (xx%) |
| Echocardiography | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| Echocardiography | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, | | | | |
| Result normal | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If abnormal, | Details | xx (xx%) | xx (xx%) | xx (xx%) |
| Orodental examination | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| Oroughtal examination | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, | | xx (xx%) | xx (xx%) | xx (xx%) |
| Result | Normal | xx (xx%) | xx (xx%) | xx (xx%) |
| Result | Abnormal | xx (xx%) | xx (xx%) | xx (xx%) |

#### 9.2.7. Concomitant treatments at inclusion

Table 21: Symptomatic or preventative treatments prescribed (safety population) at inclusion

| | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Symptomatic or preventative treatments | | | |
| prescribed in the 1st visit | | | |
| Antiemetic treatment | xx (xx%) | xx (xx%) | xx (xx%) |
| Anti-diarrheal treatment | xx (xx%) | xx (xx%) | xx (xx%) |
| Anti-neutropenic treatment | xx (xx%) | xx (xx%) | xx (xx%) |
| Anti-hypertensive treatment | xx (xx%) | xx (xx%) | xx (xx% |
| Mouthwashes and local anesthetics | xx (xx%) | xx (xx%) | xx (xx% |
| Emollients, moisturizing creams | xx (xx%) | xx (xx%) | xx (xx% |
| Analgesics | xx (xx%) | xx (xx%) | xx (xx% |
| Anti-gastro-esophageal reflux treatment | xx (xx%) | xx (xx%) | xx (xx% |
| Bisphosphonates | xx (xx%) | xx (xx%) | xx (xx% |
| Other additional anti-tumor treatment | xx (xx%) | xx (xx%) | xx (xx% |
| Details | xx (xx%) | xx (xx%) | xx (xx% |
| Other prescriptions | xx (xx%) | xx (xx%) | xx (xx%) |
| Details | xx (xx%) | xx (xx%) | xx (xx% |
| <b></b> | | | |

## 9.2.8. Supportive measures for sunitinib treatment at initiation

Table 22: Supportive measures for sunitinib treatment (safety population) at initiation

| | Call Center<br>(N=xxx) | Standard<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Information received by the patient when sunitinib treatment was started | | | |
| (several options possible) | | | |
| By the investigator him/herself | xx (xx%) | xx (xx%) | xx (xx%) |
| By the care team | xx (xx%) | xx (xx%) | xx (xx%) |
| Nurse | xx (xx%) | xx (xx%) | xx (xx%) |
| Pharmacist | xx (xx%) | xx (xx%) | xx (xx%) |
| Intern | xx (xx%) | xx (xx%) | xx (xx%) |
| CRA | xx (xx%) | xx (xx%) | xx (xx%) |
| Other | xx (xx%) | xx (xx%) | xx (xx%) |
| | xx (xx%) | xx (xx%) | xx (xx%) |
| By an information leaflet or other support/material/document given to | xx (xx%) | xx (xx%) | xx (xx%) |
| the patient | | | |
| Details of support | xx (xx%) | xx (xx%) | xx (xx%) |
| | xx (xx%) | xx (xx%) | xx (xx%) |
| Other | xx (xx%) | xx (xx%) | xx (xx%) |
| Details | xx (xx%) | xx (xx%) | xx (xx%) |
| | xx (xx%) | xx (xx%) | xx (xx%) |

## 9.3. Description of patients during the follow-up period

#### 9.3.1. Change in treatment with sunitinib (dose/dosage regimen)

Table 23: Description of changes to treatment with sunitinib in terms of dosage and dosage regimen (safety population - Call Center)

| | | Cycle 1<br>(N=xxx) | Cycle 2<br>(N=xxx) | Cycle 3<br>(N=xxx) | Cycle 4<br>(N=xxx) | Call center<br>(N=xxx) |
|---|---|---|---|---|---|---|
| At least 1 change in dose during | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| treatment with sunitinib | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Type (several options possible) | Reduction | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Increase | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| At least 1 change in dosage regiment | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| during treatment with sunitinib | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| New regimen | Details | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| - | | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Reasons for changing (patients | AE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| involved at least once for each of the | Other | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| possible reasons) | Details | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

#### 9.3.2. Tumor assessments during the follow-up period

Table 24: Tumor assessments (safety population - Call Center) during the follow-up period

| | | V1 - End of | V2 - End of cycle | V3 - End of |
|---|---|---|---|---|
| | | cycle 1 | 2 | cycle 4 |
| | | (N=xxx) | (N=xxx) | (N=xxx) |
| Tumor assessment since the last visit | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| <u>If yes,</u> | | | | |
| Radiologic investigation (several | СТ | xx (xx%) | xx (xx%) | xx (xx%) |
| options possible) | MRI | xx (xx%) | xx (xx%) | xx (xx%) |
| | PET scan | xx (xx%) | xx (xx%) | xx (xx%) |
| | radiography | xx (xx%) | xx (xx%) | xx (xx%) |
| | Ultrasound | xx (xx%) | xx (xx%) | xx (xx%) |
| Response to treatment (RECIST | CR (Complete response) | xx (xx%) | xx (xx%) | xx (xx%) |
| v1.1 criteria) | PR (Partial response) | xx (xx%) | xx (xx%) | xx (xx%) |
| | SD (Stable disease) | xx (xx%) | xx (xx%) | xx (xx%) |
| | PD (Progressive disease) | xx (xx%) | xx (xx%) | xx (xx%) |
| | NE (Not evaluable) | xx (xx%) | xx (xx%) | xx (xx%) |
| <u>If not evaluable,</u> reason | Details | xx (xx%) | xx (xx%) | xx (xx%) |

The assessment of the best response during treatment is shown in part 9.5.4., Response to treatment.

## 9.3.3. Clinical indices during the follow-up period

Table 25: Clinical indices (safety population - Call Center) during the follow-up period

| | | inclusion<br>(N=xxx) | V1 - End of<br>cycle 1<br>(N=xxx) | V2 - End of<br>cycle 2<br>(N=xxx) | V3 - End of<br>cycle 4<br>(N=xxx) |
|---|---|---|---|---|---|
| ECOG performance index assessed | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| · | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, ECOG score | 0 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 2 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 3 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 4 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Karnofsky index scored | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| <u>If yes,</u> Karnofsky index | 100% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| <del></del> | 90% - 80% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 70% - 60% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 50% - 40% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 30% - 10% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 0% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Blood pressure | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, | | | | | |
| Systolic value (mmHg) | Number<br>analyzed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Mean (±SD) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Median | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Min-Max | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Diastolic value (mmHg) | Number<br>analyzed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Mean (±SD) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Median | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Min-Max | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

# 9.3.4. Hematologic and biochemical profile during the follow-up period

Table 26: Hematologic and biochemical profile (safety population - Call Center) during the follow-up period

| | | inclusion<br>(N=xxx) | 1 | V2 - End of cycle<br>2 | V3 - End of<br>cycle 4 |
|---|---|---|---|---|---|
| | | | (N=xxx) | (N=xxx) | (N=xxx) |
| Hematologic profile | | | | | |
| Hemoglobin | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx% |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| Value (g/dL) | Number analyzed | XXX | XXX | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | XX | X |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - x |
| Neutrophils | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx% |
| • | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| Value (mm³) | Number analyzed | xxx | xxx | xxx | XXX |
| • • | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Platelets | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| Value (10 <sup>9</sup> /L) | Number analyzed | XXX | XXX | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Biochemical profile | | | | | |
| Creatinine | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| Value (mg/dL) | Number analyzed | XXX | XXX | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx | XX - XX |
| ALT (SGPT) | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| Value (U/L) | Number analyzed | xxx | XXX | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| AST (SGOT) | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

| | | inclusion<br>(N=xxx) | V1 - End of cycle<br>1<br>(N=xxx) | V2 - End of cycle<br>2<br>(N=xxx) | V3 - End of<br>cycle 4<br>(N=xxx) |
|---|---|---|---|---|---|
| If value obtained, | | | | | |
| Value (U/L) | Number analyzed | xxx | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | XX | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Calcium | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| Value (mmol/L) | Number analyzed | XXX | XXX | XXX | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | XX | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Albumin | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| Value (g/L) | Number analyzed | XXX | XXX | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| LDH | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| Value (IU/L) | Number analyzed | XXX | XXX | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |

Table 27: Abnormal values for other hematologic and biochemical indices (safety population - Call Center) during the follow-up period

| Detient in Co | II Conton group | inclusion<br>(N=xxx) | V1 - End of cycle 1 | V2 - End of cycle<br>2 | V3 - End of cycle 4 |
|---|---|---|---|---|---|
| Patient in Ca | II Center group | | (N=xxx) | (N=xxx) | (N=xxx) |
| Abnormal values for | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| biological indices | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, | | | | | |
| Hematologic profile | | | | | |
| Hematocrit | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If result abnormal, | | | | | |
| Value (in%) | Number analyzed | xxx | xxx | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |

| | | inclusion<br>(N=xxx) | V1 - End of cycle | V2 - End of cycle<br>2 | V3 - End of<br>cycle 4 |
|---|---|---|---|---|---|
| | l Center group | | (N=xxx) | (N=xxx) | (N=xxx) |
| Leucocytes | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) |
| | Not performed | ^^ (^^/) | ** (***) | ** (***) | ^^ (^^/) |
| If value obtained, | | (9/) | (9/) | /9/\ | (9/) |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If result abnormal, | | | | | |
| Value (in 10 <sup>9</sup> /L) | Number analyzed | xxx | xxx | xxx | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Biochemical profile | | | | | |
| Alkaline phosphatase | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| And the phosphatase | Value obtained Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | • | | | | |
| If value obtained,<br>abnormal result | Voc | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| aunormai resuit | Yes<br>No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | INO | XX (XXX) | XX (XXX) | XX (XXX) | XX (XXX) |
| If result abnormal, | | | | | |
| Value (in U/L) | Number analyzed | xxx | XXX | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Bilirubin | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If | | | | | |
| <u>If result abnormal,</u><br>Value (in mg/dL) | Number analyzed | xxx | xxx | xxx | XXX |
| value (III IIIg/uL) | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | XX | ×x | ×× |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| | | vo. (20%) | (.a.%) | · | vo. (vo.9/) |
| ГSH | Value obtained | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) |
| | Value not obtained<br>Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | XX (XXX) | XX (XXX) | XX (XXX) | λλ (λλλ) |
| If value obtained, | | vv. (vv%) | vv (vv%) | vv. (vv%) | w (w%) |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If result abnormal, | | | | | |
| Value (in mU/L) | Number analyzed | xxx | xxx | xxx | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| fT3 | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| · - <del>-</del> | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Marila 11 1 | , | • • | . , | | . , |
| If value obtained,<br>abnormal result | Voc | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| apnormai resuit | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | NO | | | | |
| | No | ** (***) | ** (***) | 7.0. (7.0.0°) | () |

| | | inclusion<br>(N=xxx) | V1 - End of cycle | V2 - End of cycle<br>2 | V3 - End of cycle 4 |
|---|---|---|---|---|---|
| | l Center group | | (N=xxx) | (N=xxx) | (N=xxx) |
| Value (in pmol/L) | Number analyzed | XXX | XXX | XXX | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | XX | XX | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| fT4 | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If result abnormal, | | | | | |
| Value (in pmol/L) | Number analyzed | xxx | xxx | xxx | xxx |
| value (iii pilioi) Lj | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Sodium | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If result abnormal, | | | | | |
| Value (in mmol/L) | Number analyzed | xxx | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Potassium | Value obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Value not obtained | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Not performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If value obtained, | | | | | |
| abnormal result | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| abilorillar result | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If result abnormal, | | | | | |
| Value (in mmol/L) | Number analyzed | xxx | xxx | xxx | xxx |
| - 3140 (III IIIII 01/ E/ | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | XX | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |

## $9.3.5. \ \textbf{Symptoms during the follow-up period}$

Table 28: Symptoms of patients who were followed up (safety population - Call Center) during the follow-up period

| | | V1 - End of<br>cycle 1<br>(N=xxx) | V2 - End of<br>cycle 2<br>(N=xxx) | V3 - End of<br>cycle 4<br>(N=xxx) | Overall during follow-up |
|---|---|---|---|---|---|
| Symptoms develop (several | Skin reactions or disorder | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| options possible) | Gastrointestinal disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Cardiac disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Bleeding disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Hematologic disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Infectious problems | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Pain | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Site | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | <br>Endocrine disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Inflammatory disorders (mucitis, etc.) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | General disorders (asthenia, anorexia, | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | etc.) | | | | |
| | Development of other AE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

## 9.3.6. Supportive measures during follow-up period

Table 29: Supportive measures for sunitinib treatment (safety population - call center follow-up) during the follow-up period, instituted by the doctor

| Patient in Call Center group | Start of sunitinib (N=xxx) | V1 - End of<br>cycle 1<br>(N=xxx) | V2 - End of<br>cycle 2<br>(N=xxx) | V3 - End of<br>cycle 4<br>(N=xxx) |
|---|---|---|---|---|
| Information received by the patient when treatment with | | | | |
| sunitinib was started | | | | |
| (several options possible) | | | | |
| No new information leaflet | | xx (xx%) | xx (xx%) | xx (xx%) |
| By the investigator him/herself | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| By the care team | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Nurse | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Pharmacist | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Intern | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| CRA | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Other | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| by an information leaflet or any other support/material/ | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| document given to the patient | | | | |
| Details of support | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Other | xx (xx%) | | | |
| Details | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

## 9.4. Analysis of the primary end point

Table 30: Development of AEs during the follow-up period (safety population)

| | | Number of calls<br>received < xx<br>(N=xxx) | Number of calls<br>received ≥ xx<br>(N=xxx) | Call center<br>(N=xxx) |
|---|---|---|---|---|
| At least 1 grade 3 or 4 AE whether or not related to | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| Sunitinib | | [xx; xx] | [xx; xx] | [xx; xx] |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of grade 3 or grade 4 AEs, whether or not | Number | xxx | xxx | xxx |
| related to Sunitinib per patient | analyzed | | | |
| elated to Sunitinib per patient | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Standardized grade 3 or 4 AEs, whether or not related to Sunitinib per patient, reported over the 6 months of | Number<br>analyzed | xxx | xxx | xxx |
| treatment | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| ticatilicit | • • | | , , | , , |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx |

Table 31: Description of grade 3 and 4 AEs related or unrelated to sunitinib recorded during the follow-up period (safety population)

| | | Number of calls<br>received < xx<br>(N=xxx) | Number of calls<br>received ≥ xx<br>(N=xxx) | Call center<br>(N=xxx) |
|---|---|---|---|---|
| Type of grade 3 or 4 AEs, whether or not related to | xxxx | xx (xx%) | xx (xx%) | xx (xx%) |
| Sunitinib | XXXX | xx (xx%) | xx (xx%) | xx (xx%) |
| (SOC – MedDRA category)* | xxxx | xx (xx%) | xx (xx%) | xx (xx%) |
| Type of grade 3 or 4 AEs, whether or not related to | XXXX | xx (xx%) | xx (xx%) | xx (xx%) |
| Sunitinib | xxxx | xx (xx%) | xx (xx%) | xx (xx%) |
| (PT – MedDRA category)* | xxxx | xx (xx%) | xx (xx%) | xx (xx%) |

<sup>\*</sup> Categories involving at least 2% of patients

These tables are described for patients under standard follow-up also for exploratory purposes.

## 9.5. Analysis of the secondary end points

#### 9.5.1. Sunitinib treatment

#### 9.5.1.1. Dose reductions

Table 32: Description of dose reductions (safety population)

| | | Cycle 1<br>(N=xxx) | Cycle 2<br>(N=xxx) | Cycle 3<br>(N=xxx) | Cycle 4<br>(N=xxx) | Call center<br>(N=xxx) |
|---|---|---|---|---|---|---|
| At least 1 dose reduction during | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| treatment with sunitinib | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Reason for dose reductions (patients | AE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| involved on at least 1 occasion for | Other | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| each of the possible reasons) | Details | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

The average dose reductions were xx mg/day (+/- xx).

Table 33: Dose reductions made depending on the number of calls received (safety population)

| | Number o<br>received<br>(N=xx | | | Number of calls<br>received ≥ xx<br>(N=xxx) | | Call center<br>(N=xxx) | |
|---|---|---|---|---|---|---|---|
| At least 1 dose reduction during | Yes | xx | (xx%) | xx | (xx%) | XX | (xx%) |
| treatment with sunitinib | No | xx | (xx%) | xx | (xx%) | XX | (xx%) |
| Reason for dose reductions (patients | AE | xx | (xx%) | xx | (xx%) | xx | (xx%) |
| involved on at least 1 occasion for | Other | xx | (xx%) | xx | (xx%) | XX | (xx%) |
| each of the possible reasons) | Details | XX | (xx%) | xx | (xx%) | xx | (xx%) |

## 9.5.1.2. Temporary interruptions of sunitinib treatment

Table 34: Description of temporary interruption of sunitinib treatment during the follow-up period (safety population)

| | | Cycle 1<br>(N=xxx) | Cycle 2<br>(N=xxx) | Cycle 3<br>(N=xxx) | Cycle 4<br>(N=xxx) | Call Center<br>(N=xxx) |
|---|---|---|---|---|---|---|
| At least 1 temporary interruption of | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| sunitinib treatment | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Mean duration of interruption (in days) | Number<br>analyzed | xxx | xxx | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
| Reason for interruption (patients | AE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| involved once for each of the possible | Radiotherapy | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| reasons) | Surgery | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| , | Other | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Table 35: Temporary interruption of sunitinib treatment during the follow-up period depending on number of calls received (safety population)

| | | Number of calls received < xx | Number of calls received ≥ xx | Call center<br>(N=xxx) |
|---|---|---|---|---|
| | | (N=xxx) | (N=xxx) | |
| At least 1 temporary interruption of | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| sunitinib treatment | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Reason for interruption (patients | AE | xx (xx%) | xx (xx%) | xx (xx%) |
| involved once for each of the possible | Radiotherapy | xx (xx%) | xx (xx%) | xx (xx%) |
| reasons) | Surgery | xx (xx%) | xx (xx%) | xx (xx%) |
| | Other | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details | xx (xx%) | xx (xx%) | xx (xx%) |

#### 9.5.1.3. Discontinuation of sunitinib treatment

Table 36: Description of discontinuations of sunitinib treatment during the follow-up period (safety population)

| | | Number of calls | Number of calls | Call center |
|---|---|---|---|---|
| | | received < xx | received ≥ xx | (N=xxx) |
| | | (N=xxx) | (N=xxx) | |
| Patients who stopped sunitinib | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Reason for stopping sunitinib | Progressive disease | xx (xx%) | xx (xx%) | xx (xx%) |
| | Toxicity | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details | xx (xx%) | xx (xx%) | xx (xx%) |
| | Intercurrent disease | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details | 2 | xx (xx%)xx (xx%) | x <b>x</b> x( <b>1111111111111</b> |
| | Patient choice | xx (xx%) | xx (xx%) | xx (xx%) |
| | Doctor choice | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details | xx (xx%) | xx (xx%) | xx (xx%) |
| | Died | xx (xx%) | xx (xx%) | xx (xx%) |
| | Other | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of cycles before | 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| discontinuation | 2 | xx (xx%) | xx (xx%) | xx (xx%) |
| | 3 | xx (xx%) | xx (xx%) | xx (xx%) |
| | 4 | xx (xx%) | xx (xx%) | xx (xx%) |
| Duration of treatment (months) | Number analyzed | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Duration of treatment if stopped | Number analyzed | xxx | xxx | xxx |
| (months) | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx |

# 9.5.2. Number of unpredicted medical procedures either related or unrelated to sunitinib

Table 37: Requirements for medical procedures by cycle during the follow-up period (safety population)

| | | V1 - End of<br>cycle 1<br>(N=xxx) | V2 - End of<br>cycle 2<br>(N=xxx) | V3 - End of<br>cycle 4<br>(N=xxx) | Call Center<br>(N=xxx) |
|---|---|---|---|---|---|
| At least 1 consultation | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, at least 1 | Planned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| , | Unplanned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| At least 1 hospitalization | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| · | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, at least 1 | Planned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| , . | Unplanned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| At least 1 hospitalization and | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 consultation | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| At least 1 call to a health | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| professional | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, at least 1 | Planned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Unplanned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Table 38: Number of medical procedures per cycle during the follow-up period (safety population)

| | | V1 - End of | V2 - End of | V3 - End of | |
|---|---|---|---|---|---|
| | | cycle 1 | cycle 2 | cycle 4 | <b>Call Center</b> |
| Subject to sufficient numbers | | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| Requirement for consultations | | | | | |
| Number of planned consultations performed per cycle | Number | xxx | xxx | xxx | xxx |
| | analyzed | | | | |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Number of unpredicted consultations performed per | Number | xxx | xxx | xxx | xxx |
| cycle | analyzed | | | | |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Total number of consultations performed per cycle | Number | xxx | xxx | xxx | xxx |
| | analyzed | | | | |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Requirement for hospitalizations | | | | | |
| Number of planned hospitalizations performed per | Number | XXX | XXX | XXX | xxx |
| <u>cycle</u> | analyzed | | | | |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Total number of hospitalizations performed per cycle | Number | xxx | xxx | xxx | xxx |
| | analyzed | | | | |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |

| Subject to sufficient numbers | | V1 - End of<br>cycle 1<br>(N=xxx) | V2 - End of<br>cycle 2<br>(N=xxx) | V3 - End of<br>cycle 4<br>(N=xxx) | Call Center<br>(N=xxx) |
|---|---|---|---|---|---|
| Number of planned consultations and hospitalizations | Number | xxx | xxx | xxx | xxx |
| performed <u>per cycle</u> | analyzed | | | | |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Requirement for consultations AND hospitalizations | | | | | |
| Number of planned consultations AND hospitalizations performed per cycle | Number<br>analyzed | xxx | xxx | xxx | xxx |
| performed <u>per cycle</u> | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Total number of consultations AND hospitalizations performed per cycle | Number<br>analyzed | xxx | xxx | xxx | xxx |
| periorimed <u>per cycle</u> | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Total number of consultations AND hospitalizations performed per cycle | Number<br>analyzed | xxx | xxx | xxx | xxx |
| performed <u>per cycle</u> | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | ×x | ×× |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Requirement for calls to a health professional | | | | | |
| Total number of planned calls made <u>per cycle</u> | Number<br>analyzed | XXX | XXX | XXX | XXX |
| | ,<br>Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | XX | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Number of unplanned calls made <u>per cycle</u> | Number<br>analyzed | xxx | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |
| Total number of calls made <u>per cycle</u> | Number<br>analyzed | xxx | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx |

#### 9.5.3. Adherence to treatment

Table 39: Morisky scale items during the follow-up period (safety population)

| | | End of cycle 1<br>(N=xxx) | End of cycle 2<br>(N=xxx) | End of cycle<br>4<br>(N=xxx) |
|---|---|---|---|---|
| Morisky questionnaire items | | | | • |
| Has already forgotten to take treatment | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| , • | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Occasionally has difficulty remembering to take | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| treatment | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Occasionally stops taking treatment when he/she feels | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| better | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Occasionally stops taking treatment when he/she feels | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| less well | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Additional question about the AEs | | | | |
| Occasionally reduced or adjusts treatment when an | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| adverse event develops | No | xx (xx%) | xx (xx%) | xx (xx%) |

Table 40: Assessment of adherence during the follow-up period (safety population)

| | | End of cycle 1<br>(N=xxx) | End of cycle 2<br>(N=xxx) | End of cycle<br>4<br>(N=xxx) |
|---|---|---|---|---|
| MMAS-4 score (adherence score)* | Number analyzed | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | xx | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Level of adherence | High: 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Mean: 1 or 2 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Low: 3 or 4 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Missing value | xx - | xx - | xx - |
| "Adherent" patient | Yes: 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| · | No: >=1 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Missing value | xx - | xx - | xx - |
| Difference in adherence score | Number analyzed | - | - | XXX |
| between the end of C1 and C4 | Mean (±SD) | - | - | xx (± xx) |
| | Median | - | - | XX |
| | Min-Max | - | - | xx - x |
| Difference in adherence score | Improvement | - | - | xx (xx%) |
| between the end of C1 and C4 | Stable score | - | - | xx (xx%) |
| | Deterioration | - | - | xx (xx%) |
| | Missing value | - | - | xx - |

<sup>\*</sup> From 0 to 4: a low score represents improved adherence.

# • Assessment of adherence in week 4 of cycles 1, 2 and 4 by telephone in patients in the CC arm

Table 41: Morisky scale items in week 4 of cycles 1, 2 and 4 (safety population)

| Carried out by telephone | | Call, W4<br>cycle 1<br>(N=xxx) | Call, W4<br>cycle 2<br>(N=xxx) | Call, W4<br>cycle 4<br>(N=xxx) |
|---|---|---|---|---|
| Morisky questionnaire items: | | | | |
| Has already forgotten to take treatment | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Occasionally has difficulty remembering to take | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| treatment | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Occasionally stops taking treatment when he/she feels | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| better | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Occasionally stops taking treatment when he/she feels | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| less well | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Additional guestion about the AE | | | | |
| Occasionally reduced or adjusts treatment when an | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| adverse event develops | No | xx (xx%) | xx (xx%) | xx (xx%) |

Table 42: Assessment of adherence in week 4 of cycles 1, 2 and 4 (safety population)

| Carried out by telep | hone | Call, W4<br>cycle 1<br>(N=xxx) | Call, W4<br>cycle 2<br>(N=xxx) | Call, W4<br>cycle 4<br>(N=xxx) |
|---|---|---|---|---|
| MMAS-4 score (adherence score)* | Number analyzed | xxx | xxx | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | xx | X |
| | Min-Max | xx - xx | xx - xx | xx - x |
| Level of adherence | High: 0 | xx (xx%) | xx (xx%) | xx (xx% |
| | Moderate: 1 or 2 | xx (xx%) | xx (xx%) | xx (xx% |
| | Low: 3 or 4 | xx (xx%) | xx (xx%) | xx (xx% |
| | Missing value | xx - | xx - | xx |
| "Adherent" patient | Yes: 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| • | No: >=1 | xx (xx%) | xx (xx%) | xx (xx% |
| | Missing value | xx - | xx - | xx · |

From 0 to 4: a low score represents improved adherence.

Table 43: Consistency between assessment of adherence at W4 (telephone) and W6 (self-completed questionnaire) in each cycle 1, 2 and 4 (safety population)

| | | | herence at W6 (M<br>eted paper questi | • | Coefficient<br>Kappa |
|---|---|---|---|---|---|
| Cycle 1 | | High: | Moderate: | Low: | карра |
| | | 0<br>(N=xxx) | 1 or 2<br>(N=xxx) | 3 or 4<br>(N=xxx) | |
| Level of adherence at W4 (MMAS-4) | High: 0 | xx (xx%) | xx (xx%) | xx (xx%) | xx |
| (telephone) | Moderate: 1 or 2 | xx (xx%) | xx (xx%) | xx (xx%) | |
| ` ' ' | Low: 3 or 4 | xx (xx%) | xx (xx%) | xx (xx%) | |
| | Missing value | xx - | xx - | xx - | |
| | | Level of ad | herence at W6 (M | MAS-4) | Coefficient |
| | | Self-comple | eted paper questi | onnaire | Карра |
| Cycle 2 | | High: | Moderate: | Low: | |
| | | 0 | 1 or 2 | 3 or 4 | |
| | | (N=xxx) | (N=xxx) | (N=xxx) | |
| Level of adherence at W4 (MMAS-4) | High: 0 | xx (xx%) | xx (xx%) | xx (xx%) | xx |
| (telephone) | Moderate: 1 or 2 | xx (xx%) | xx (xx%) | xx (xx%) | |
| | Low: 3 or 4 | xx (xx%) | xx (xx%) | xx (xx%) | |
| | Missing value | xx - | xx - | xx - | |
| | | Level of ad | herence at W6 (M | MAS-4) | Coefficient |
| | | Self-comple | eted paper questi | onnaire | Карра |
| Cycle 4 | | High: | Moderate: | Low: | |
| | | 0 | 1 or 2 | 3 or 4 | |
| | | (N=xxx) | (N=xxx) | (N=xxx) | |
| Level of adherence at W4 (MMAS-4) | High: 0 | xx (xx%) | xx (xx%) | xx (xx%) | xx |
| (telephone) | Moderate: 1 or 2 | xx (xx%) | xx (xx%) | xx (xx%) | |
| | Low: 3 or 4 | xx (xx%) | xx (xx%) | xx (xx%) | |
| | Missing value | xx - | xx - | xx - | |

## 9.5.4. Response to the sunitinib treatment

Table 44: Response to sunitinib treatment (FAS population)

| | | Number of calls<br>received < xx<br>(N=xxx) | Number of calls<br>received ≥ xx<br>(N=xxx) | Call center<br>(N=xxx) |
|---|---|---|---|---|
| Best response obtained during | CR (Complete response) | xx (xx%) | xx (xx%) | xx (xx%) |
| treatment according to RECIST v1.1 | PR (Partial response) | xx (xx%) | xx (xx%) | xx (xx%) |
| criteria | SD (Stable disease) | xx (xx%) | xx (xx%) | xx (xx%) |
| | PD (Progressive disease) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Missing value | xx - | xx - | xx - |
| Best complete or partial response | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| (Objective response rate) | No | xx (xx%) | xx (xx%) | xx (xx%) |
| | Missing value | xx - | xx - | xx - |

#### 9.5.5. Patient support

#### 9.5.5.1. Number of calls

Table 45: Frequency of calls made during sunitinib treatment by cycle and overall (FAS population)

| | | Patier | ts per sunitir | ib treatment | cycle | Total |
|---|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 | (N=xxx) |
| | | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | |
| Number of <u>planned</u> completed calls per patient | Number<br>analyzed | xxx | xxx | xxx | xxx | xxx |
| • | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
| Number of <u>unplanned</u> completed calls per patient | Number<br>analyzed | xxx | xxx | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |
| Total number of completed calls per patient | Number<br>analyzed | xxx | xxx | xxx | xxx | xxx |
| parameter 1 | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | xx | xx | xx | xx | xx |
| | Min-Max | xx - xx | xx - xx | xx - xx | xx - xx | xx - xx |

#### 9.5.5.2. Actions by doctors and patients

Table 46: Actions by doctors and patients assessed during the first call (FAS population)

| ccording to the patient, at the time of the first call: | | 1 <sup>st</sup> Call<br>(N=xxx) |
|---|---|---|
| ction by doctor | | |
| The doctor clearly explained how to take the treatment | Yes | xx (xx% |
| | No | xx (xx% |
| The patient was given documentation about the treatment by | Yes, information leaflet | xx (xx% |
| the doctor or medical team | Yes, Sutent® diary | xx (xx% |
| | No | xx (xx |
| The doctor explained how to manage any side effects due to | Yes | xx (xx |
| treatment which could occur | No | xx (xx |
| Prescriptions or orders for supportive medical treatments by | Yes | xx (xx |
| the doctor | No | xx (xx |
| ction by patient | | |
| Sutent® taken | Yes | xx (xx |
| | No | xx (xx |
| If no, reason | Forgot to start | xx (xx |
| | Stressed/worried about the idea of taking | xx (xx |
| | the drug | |
| | Other reason | xx (xx |
| | Details | |

Table 47: Actions by doctors and patients assessed during the first call in cycles 2, 3 and 4 (FAS population)

| According to the patient, at the time of the first call | in cycles 2, 3 and 4: | 1 <sup>st</sup> call,<br>cycle 2<br>(N=xxx) | 1 <sup>st</sup> call,<br>cycle 3<br>(N=xxx) | 1 <sup>st</sup> call,<br>cycle 4<br>(N=xxx) |
|---|---|---|---|---|
| Actions by patient | | , , | , , | , , |
| A new cycle of Sutent® was due to be started: | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| restarted Sutent® | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If no, reason | Planned restart | xx (xx%) | xx (xx%) | xx (xx%) |
| | Forgot to restart | xx (xx%) | xx (xx%) | xx (xx%) |
| | Stressed/worried about the idea of taking the drug | xx (xx%) | xx (xx%) | xx (xx%) |
| | Development of an AE | xx (xx%) | xx (xx%) | xx (xx%) |
| | Treatment delayed or interrupted temporarily by the doctor | xx (xx%) | xx (xx%) | xx (xx%) |
| | Other reason | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details | xx (xx%) | xx (xx%) | xx (xx%) |
| Action by doctor | | | | |
| Dose and/or dosage regimen amended by the | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| doctor in the last visit | No | xx (xx%) | xx (xx%) | xx (xx%) |
| Prescription or order for supportive medicinal | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| products by the doctor | No | xx (xx%) | xx (xx%) | xx (xx%) |

#### 9.5.5.3. Advice delivered

Table 48: Advice given during calls by the support call center by cycle and overall (FAS population)

| | N=Patie | nts who were | called at lea | st once | Total Patients |
|---|---|---|---|---|---|
| Advice delivered during calls (several options possible) | Cycle 1<br>(N=xxx) | Cycle 2<br>(N=xxx) | Cycle 3<br>(N=xxx) | Cycle 4<br>(N=xxx) | (N=xxx) |
| Advice about managing the treatment | | | | | |
| Advice about taking Sutent® | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Advice about using the Sutent® follow-up diary | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Reporting any AE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| General preventative advice | | | | | |
| Advice about taking preventative systemic treatments | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Lifestyle advice | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Food/dietetic advice | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Oro-dental hygiene advice | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Specific preventative advice for a type of AE | | | | | |
| Prevention of skin toxicities | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Prevention of gastrointestinal disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Prevention of cardiac disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Prevention of infectious/inflammatory problems | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Other preventative advice | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Actions recommended to patient | | | | | |
| Do not forget the planned consultation with the oncologist | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Get the additional investigations requested performed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

#### 9.5.6. Satisfaction with the call center

#### 9.5.6.1. Doctors' satisfaction with the call center

Table 49: Satisfaction of doctors who included patients followed up by the call center with the patient treatment management call center

| | | Doctors<br>who included at least 1<br>patient into the Call Cente<br>arm |
|---|---|---|
| Satisfaction assessed at the end of the patient follow-up period | | (N=xxx) |
| Satisfaction with the advice | | |
| - In terms of the reduction in the number and/or frequency of | Very satisfied | xx (xx% |
| grade 3/4 AEs as a result of the advice delivered during the | Satisfied | xx (xx% |
| support process | Not particularly | xx (xx% |
| | satisfied | ya. (ya.9) |
| | Not satisfied | xx (xx% |
| | No opinion | xx (xx% |
| - With the improvement in adherence to treatment through the | Very satisfied | xx (xx% |
| support | Satisfied | xx (xx% |
| | Not particularly | xx (xx% |
| | satisfied | |
| | Not satisfied | xx (xx% |
| | No opinion | xx (xx% |
| - With the change in patient's quality of life through the advice | Very satisfied | xx (xx% |
| delivered by the call center | Satisfied | xx (xx% |
| delivered by the call center | Not particularly | xx (xx% |
| | satisfied | |
| | Not satisfied | xx (xx% |
| | No opinion | xx (xx% |
| Satisfaction with care | | |
| - Feeling that the treatment management call center care reduced | Very satisfied | xx (xx% |
| workload | Satisfied | xx (xx% |
| | Not particularly | xx (xx% |
| | satisfied | |
| | Not satisfied | xx (xx% |
| | No opinion | xx (xx% |
| Overall satisfaction of patient care with the call center | Very satisfied | xx (xx% |
| | Satisfied | xx (xx% |
| | Not particularly | xx (xx% |
| | satisfied | |
| | Not satisfied | xx (xx% |
| | No opinion | xx (xx% |
| Overall satisfaction: Doctor "satisfied" or "very satisfied" | Yes | xx (xx% |
| | No | xx (xx% |
| Desire to continue this type of support | Yes | xx (xx% |
| , | No | xx (xx% |

A 3 axis radar plot shows the mean satisfaction scores for each dimension. The area of the polygon and percentage surface area covered are shown on the plot. A high represents greater general satisfaction.

Table 50: Characteristics of doctors who were satisfied or very satisfied with the support from the patient treatment management call center

| | | Overall satisfied or very satisfied with the<br>support | |
|---|---|---|---|
| | | Yes | No |
| | | (N=xxx) | (N=xxx) |
| Age of doctor | Number analyzed | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) |
| | Median | xx | xx |
| | Min-Max | xx - xx | xx - xx |
| Sex | Male | xx (xx%) | xx (xx%) |
| | Female | xx (xx%) | xx (xx%) |
| Number of patients who used the call center | Number analyzed | xxx | xxx |
| for at least 50% of the planned calls | Mean (±SD) | xx (± xx) | xx (± xx) |
| · | Median | xx | xx |
| | Min-Max | xx - xx | xx - xx |
| Average number of planned and unplanned | Number analyzed | xxx | xxx |
| calls received by the patients | Mean (±SD) | xx (± xx) | xx (± xx) |
| | Median | xx | xx |
| | Min-Max | xx - xx | xx - xx |

#### 9.5.6.2. Patient satisfaction with the call center

Table 51: Satisfaction of patients included in the Call Center arm with the call center (FAS Call Center population)

| Patient satisfaction assessed at the end of their follow-up in the study (end of cycle 4 or end of treatment) | | Total<br>(N=xxx) |
|---|---|---|
| Satisfaction with the advice | | |
| - With the preventative advice given to avoid sunitinib related | Very satisfied | xx (xx |
| complications | Satisfied | xx (xx |
| | Not particularly satisfied | xx (xx |
| | Not satisfied | xx (xx |
| | No opinion | xx (xx |
| - With the advice given to reduce/resolve side effects due to | Very satisfied | xx (xx |
| sunitinib | Satisfied | xx (xx |
| | Not particularly satisfied | xx (xx |
| | Not satisfied | xx (xx |
| | No opinion | xx (xx |
| Natish the conscitut of the call contact to divert the notices to a | Voncentiation | xx (xx |
| - With the capacity of the call center to direct the patient to a | Very satisfied | xx (xx |
| general practitioner/oncologist when the situation required this | Satisfied | xx (xx |
| | Not particularly satisfied Not satisfied | xx (xx |
| | No opinion | xx (xx |
| | νο ομιποπ | ( |
| Satisfaction with care | | ( |
| - With the explanations given about the disease, treatment | Very satisfied | xx (xx |
| and/or their side effects | Satisfied | xx (xx |
| | Not particularly satisfied | xx (xx |
| | Not satisfied | xx (xx<br>xx (xx |
| | No opinion | ** (** |
| Satisfaction with the service | | |
| <ul> <li>With the response given to questions, problems and/or</li> </ul> | Very satisfied | xx (xx |
| about the patient him/herself | Satisfied | xx (xx |
| | Not particularly satisfied | xx (xx |
| | Not satisfied | xx (xx |
| | No opinion | xx (xx |
| - With the frequency and duration of calls received from the | Very satisfied | xx (xx |
| patient's perspective | Satisfied | xx (xx |
| | Not particularly satisfied | xx (xx |
| | Not satisfied | xx (xx |
| | No opinion | xx (xx |
| - Availability of nurses from the call center through the toll | Very satisfied | xx (xx |
| free number available | Satisfied | xx (xx |
| | Not particularly satisfied | xx (xx |
| | Not satisfied | xx (xx |
| | No opinion | xx (xx |
| Overall satisfaction with support in management of sunitinib | Very satisfied | xx (xx |
| treatment | Satisfied | xx (xx |
| treatment | Not particularly satisfied | xx (xx |
| | Not satisfied | xx (xx |
| | No opinion | xx (xx |
| Overall satisfaction: Patient "satisfied" or "very satisfied" | · | xx (xx |
| Overall satisfaction: Patient "satisfied" or "very satisfied" | Yes | xx (xx |

A 4 axes radar plot simultaneously shows the mean scores for each satisfaction dimension. The area of the polygon and percentage of the surface area covered will be shown on this plot. A higher area represents greater general satisfaction.

Table 52: Other satisfaction indicators for patients included in the Call Center arm with the call center (FAS Call Center population)

| Satisfaction assessed at the end of the final visit at 6 weeks in cycle 4 or in the treatment | | Total<br>(N=xxx) |
|---|---|---|
| discontinuation visit | | |
| Desire to continue this type of support | Yes, completely | xx (xx%) |
| ,, ., | Possibly | xx (xx%) |
| | Not really | xx (xx%) |
| | Not at all | xx (xx%) |
| | No opinion | xx (xx%) |
| Liable to recommend this type of follow-up to a member of | Yes, completely | xx (xx%) |
| the family circle | Possibly | xx (xx%) |
| , | Not really | xx (xx%) |
| | Not at all | xx (xx%) |
| | No opinion | xx (xx%) |
| Need experienced during the study for actions proposed by | Yes | xx (xx%) |
| the call center | No | xx (xx%) |

The comments given by patients in the self-completed satisfaction questionnaires will also be provided in this section.
Table 53: Characteristics of patients who were satisfied or very satisfied with the support, in patients in the Call Center arm (FAS Call Center population)

| | | Overall very satisfied or very satisfied with the support | |
|---|---|---|---|
| | | Yes<br>(N=xxx) | No<br>(N=xxx) |
| Characteristics at inclusion | | | |
| Age (years) | Number analyzed | XXX | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) |
| | Median | XX | xx |
| | Min-Max | xx - xx | xx - xx |
| Sex | Male | xx (xx%) | xx (xx%) |
| | Female | xx (xx%) | xx (xx%) |
| ECOG score | 0 | xx (xx%) | xx (xx%) |
| | 1 | xx (xx%) | xx (xx%) |
| | 2 | xx (xx%) | xx (xx%) |
| | 3 | xx (xx%) | xx (xx%) |
| | 4 | xx (xx%) | xx (xx%) |
| | Not stated | | |
| Risk score – Heng et al. criteria | Good | xx (xx%) | xx (xx%) |
| <b>0</b> | Intermediary | xx (xx%) | xx (xx%) |
| | Poor | xx (xx%) | xx (xx%) |
| | Not available | xx (xx%) | xx (xx%) |
| Fuhrman grade | I | xx (xx%) | xx (xx%) |
| · · | II | xx (xx%) | xx (xx%) |
| | III | xx (xx%) | xx (xx%) |
| | IV | xx (xx%) | xx (xx%) |
| Metastatic renal cell carcinoma grade | Yes | xx (xx%) | xx (xx%) |
| <b>G</b> | No | xx (xx%) | xx (xx%) |
| Previous or current comorbidities | Yes | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) |
| Concomitant treatment | Yes | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) |
| Characteristics during the follow-up | | | |
| <u>period</u> | | | |
| Number of calls achieved | Number analyzed | XXX | XXX |
| | Mean (±SD) | xx (± xx) | xx (± xx) |
| | Median<br>Min-Max | xx<br>xx - xx | xx<br>xx - xx |
| Development of AEs | Yes | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) |
| Development of grade 3/4 AEs | Yes | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) |

## 9.6. Pharmacovigilance

Note: The pharmacovigilance analysis will be described both according to severity (AE/SAE) and overall.

Table 54: Description of all of the AEs declared during the study (Safety population)

| | | Safety popula<br>(N=xxx) | ation |
|---|---|---|---|
| Type of AEs (SOC – MedDRA category)* | xxxx | xx | (xx% |
| | xxxx | xx | (xx% |
| | XXXX | XX | (xx% |
| Гуре of AEs | xxxx | XX | (xx% |
| (PT – MedDRA category)* | XXXX | xx | (xx% |
| | XXXX | XX | (xx% |
| cycle | cycle 1 | xx | (xx% |
| | cycle 2 | XX | (xx% |
| | cycle 3 | xx | (xx% |
| | cycle 4 | XX | (xx% |
| Severity | Non-serious | xx | (xx% |
| | Serious | XX | (xx% |
| If serious, severity criteria | Fatal | xx | (xx% |
| | Life-threatening | xx | (xx% |
| | Hospitalization/prolongation of | xx | (xx% |
| | hospitalization | | |
| | Congenital abnormality/ malformation | xx | (xx% |
| | Permanent or severe invalidity/ | XX | (xx% |
| | incapacity Significant medical event | xx | (xx% |
| Grade | 1 | xx | (xx% |
| 5.440 | 2 | | `<br>(xx% |
| | 3 | | `<br>(xx% |
| | 4 | | (xx% |
| | 5 | | (xx% |
| | Not applicable | | (xx% |
| Causality of the AEs with sunitinib | Related to administration of Sutent® | xx | (xx% |
| | Related to a concomitant medicinal product | xx | (xx% |
| | Related to Sutent and another concomitant medicinal product | xx | (xx% |
| | Related neither to Sutent nor another | xx | (xx% |
| | medicinal product | *** | (7000 |
| | Unknown | XX | (xx% |
| Outcome | Recovered | xx | (xx% |
| | Recovered with sequelae | xx | (xx% |
| | Currently recovering | xx | (xx% |
| | Not recovered | xx | (xx% |
| | Unknown | XX | (xx% |
| Corrective medical action | Prescription of a treatment | | (xx% |
| | Medical consultation | | (xx% |
| | Hospitalization | | (xx% |
| | Other | xx | (xx% |
| | Not applicable | xx | (xx% |
| Last action undertaken for Sutent during the AE | Discontinuation (temporary or permanent, or dose delayed) | xx | (xx% |
| | Increased dosage | xx | (xx% |
| | Reduced dosage | xx | (xx% |

| | | Safety population<br>(N=xxx) |
|---|---|---|
| | Change in dosage regimen | xx (xx%) |
| | Unknown | xx (xx%) |
| | Not applicable | xx (xx%) |
| Specific situation | No specific situation | xx (xx%) |
| • | Exposure during pregnancy | xx (xx%) |
| | Overdose | xx (xx%) |
| | Medication error/Risk of medication | xx (xx%) |
| | error | |
| | Exposure during breast-feeding | xx (xx%) |
| | Misuse | xx (xx%) |
| | Lack of efficacy | xx (xx%) |
| | Off-label use | xx (xx%) |
| | Extravasation | xx (xx%) |
| | Occupational exposure | xx (xx%) |

<sup>\*</sup> Categories involving at least 2% of patients

Table 55: Description of all AEs related to sunitinib declared during the follow-up period (Safety population)

| AEs related to sunitinib* | | Safety population (N=xxx) | n |
|---|---|---|---|
| Type of AE (SOC – MedDRA category)** | XXXX | xx (xx | x%) |
| | xxxx | xx (xx | x%) |
| | xxxx | xx (xx | x%) |
| Type of AE | xxxx | xx (xx | • |
| (PT – MedDRA category)** | XXXX | xx (xx | |
| | xxxx | xx (xx | x%) |
| Cycle | cycle 1 | xx (xx | |
| | cycle 2 | xx (xx | |
| | cycle 3 | xx (xx | |
| | cycle 4 | xx (xx | x%) |
| Severity | Non-serious | xx (xx | x%] |
| | Serious | xx (xx | x%] |
| If serious, severity criteria | Fatal | xx (xx | |
| | Life-threatening | xx (xx | x% |
| | Hospitalization/prolongation of hospitalization | xx (xx | x% |
| | Congenital abnormality/ malformation | xx (xx | x% |
| | Permanent or severe invalidity/ incapacity | xx (xx | х% |
| | Significant medical event | xx (xx | x% |
| Grade | 1 | xx (xx | x% |
| | 2 | xx (xx | x% |
| | 3 | xx (xx | x%] |
| | 4 | xx (xx | x%] |
| | 5 | xx (xx | x%] |
| | Not applicable | xx (xx | x%] |
| Causality of the AEs with sunitinib | Related to administration of Sutent® | xx (xx | x%` |
| Causanty of the ALS with summing | Related to a concomitant medicinal | xx (xx | |
| | product | | |
| | Related to Sutent and another | xx (xx | x%] |
| | concomitant medicinal product | | |
| | Related neither to Sutent nor another medicinal product | xx (xx | x%] |
| | Unknown | xx (xx | x%] |
| Outcome | Recovered | xx (xx | x% |

| AEs related to sunitinib* | | Safety population<br>(N=xxx) |
|---|---|---|
| | Recovered with sequelae | xx (xx%) |
| | Currently recovering | xx (xx%) |
| | Not recovered | xx (xx%) |
| | Unknown | xx (xx%) |
| Corrective medical action | Prescription of a treatment | xx (xx%) |
| | Medical consultation | xx (xx%) |
| | Hospitalization | xx (xx%) |
| | Other | xx (xx%) |
| | Not applicable | xx (xx%) |
| Last action undertaken for Sutent during the AE | Discontinuation (temporary or permanent, or dose delayed) | xx (xx%) |
| | Increased dosage | xx (xx%) |
| | Reduced dosage | xx (xx%) |
| | Unchanged dosage | xx (xx%) |
| | Change in dosage regimen | xx (xx%) |
| | Unknown | xx (xx%) |
| | Not applicable | xx (xx%) |
| Specific situation | No specific situation | xx (xx%) |
| | Exposure during pregnancy | xx (xx%) |
| | Overdose | xx (xx%) |
| | Medication error/Risk of medication error | xx (xx%) |
| | Exposure during breast-feeding | xx (xx%) |
| | Misuse | xx (xx%) |
| | Lack of efficacy | xx (xx%) |
| | Off-label use | xx (xx%) |
| | Extravasation | xx (xx%) |
| | Occupational exposure | xx (xx%) |

<sup>\*</sup> AE related to sunitinib if the relationship is entered as "Related to taking Sutent®" or "Related to Sutent® and another concomitant medicinal product".

<sup>\*\*</sup> Categories involving at least 2% of patients

## 9.7. Supplementary analysis: Patient follow-up "Standard follow-up"

## 9.7.1. Tumor assessment during the follow-up period

Table 56: Tumor assessments (safety population- standard follow-up) during the follow-up period

| | | V1 - End of | V2 - End of cycle | V3 - End of |
|---|---|---|---|---|
| | | cycle 1 | 2 | cycle 4 |
| | | (N=xxx) | (N=xxx) | (N=xxx) |
| Tumor assessment since the last visit | Yes | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, | | | | |
| Radiologic investigation (several | CT | xx (xx%) | xx (xx%) | xx (xx%) |
| possible options) | MRI | xx (xx%) | xx (xx%) | xx (xx%) |
| | PET scan | xx (xx%) | xx (xx%) | xx (xx%) |
| | Radiography | xx (xx%) | xx (xx%) | xx (xx%) |
| | Ultrasound | xx (xx%) | xx (xx%) | xx (xx%) |
| Response to treatment (RECIST | CR (Complete response) | xx (xx%) | xx (xx%) | xx (xx%) |
| v1.1 criteria) | PR (Partial response) | xx (xx%) | xx (xx%) | xx (xx%) |
| | SD (Stable disease) | xx (xx%) | xx (xx%) | xx (xx%) |
| | PD (Progression) | xx (xx%) | xx (xx%) | xx (xx%) |
| | NE (Not evaluable) | xx (xx%) | xx (xx%) | xx (xx%) |
| If <u>not evaluable,</u> reason | Details | xx (xx%) | xx (xx%) | xx (xx%) |

## 9.7.2. Clinical indices during the follow-up period

Table 57: Clinical indices (safety population- standard follow-up) during the follow-up period

| | | inclusion | V1 - End of | V2 - End of | V3 - End of |
|---|---|---|---|---|---|
| | | (N=xxx) | cycle 1<br>(N=xxx) | cycle 2<br>(N=xxx) | cycle 4<br>(N=xxx) |
| ECOG performance index assessed | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| · | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, ECOG score | 0 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| - | 1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 2 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 3 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 4 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Karnofsky index scored | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, Karnofsky index | 100% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 90% - 80% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 70% - 60% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 50% - 40% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 30% - 10% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | 0% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Blood pressure | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

| | | inclusion<br>(N=xxx) | V1 - End of<br>cycle 1<br>(N=xxx) | V2 - End of<br>cycle 2<br>(N=xxx) | V3 - End of<br>cycle 4<br>(N=xxx) |
|---|---|---|---|---|---|
| If yes, | | | | | |
| Systolic value (mmHg) | Number<br>analyzed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Mean (±SD) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Median | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Min-Max | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Diastolic value (mmHg) | Number<br>analyzed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Mean (±SD) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Median | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Min-Max | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

### 9.7.3. Symptoms during the follow-up period

Table 58: Symptoms (safety population- standard follow-up) during the follow-up period

| | | V1 - End of<br>cycle 1<br>(N=xxx) | V2 - End of<br>cycle 2<br>(N=xxx) | V3 - End of<br>cycle 4<br>(N=xxx) | Overall during follow-up |
|---|---|---|---|---|---|
| Symptoms develop (several | Skin reactions or disorder | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| options possible) | Gastrointestinal disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Cardiac disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Bleeding disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Hematologic disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Infectious problems | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Pain . | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Site | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Details | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | <br>Endocrine disorders | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx% |
| | Inflammatory disorders (mucitis, etc.) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | General disorders (asthenia, anorexia, | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx% |
| | etc.) | | | | |
| | Development of other AE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx% |
| | Details | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx% |

### 9.7.4. Supportive measures during the follow-up period

Table 59: Supportive measures for sunitinib treatment (safety population- standard follow-up) during the follow-up period, instituted by the doctor

| | Start of<br>sunitinib<br>(N=xxx) | V1 - End of<br>cycle 1<br>(N=xxx) | V2 - End of<br>cycle 2<br>(N=xxx) | V3 - End of<br>cycle 4<br>(N=xxx) |
|---|---|---|---|---|
| Information received by the patient when treatment with | | | | |
| sunitinib was started | | | | |
| (several options possible) | | | | |
| No new information leaflet | | xx (xx%) | xx (xx%) | xx (xx%) |
| By the investigator him/herself | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| By the care team | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Nurse | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Pharmacist | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Intern | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| CRA | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Other | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| By an information leaflet or any other support/materials/ | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| document given to the patient | | | | |
| Details of the support | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Other | xx (xx%) | | | |
| Details | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

## 9.7.5. Study criteria

Table 60: Follow-up data (safety population- standard follow-up)

| | | Standard<br>follow-up<br>(N=xxx) |
|---|---|---|
| At least 1 grade 3 or 4 AE whether or not related to | Yes | xx (xx%) |
| Sunitinib | No | xx (xx%) |
| At least 1 dose reduction during treatment with sunitinib | Yes | xx (xx%) |
| | No | xx (xx%) |
| Reason for dose reductions (patients involved on at least 1 occasion for each of the possible reasons) | AE | xx (xx%) |
| | Other | xx (xx%) |
| | Details | xx (xx%) |
| At least 1 temporary interruption of sunitinib | Yes | xx (xx%) |
| · · · · | No | xx (xx%) |
| Reason for interruption (patients involved once for each of the possible reasons) | AE | xx (xx%) |
| | Radiotherapy | xx (xx%) |
| | Surgery | xx (xx%) |
| | Other | |
| | Details | |
| Best response obtained during treatment | CR (Complete response) | xx (xx%) |
| | PR (Partial response) | xx (xx%) |
| | SD (Stable disease) | xx (xx%) |
| | PD (Progressive disease) | xx (xx%) |
| | Missing value | xx<br>- |
| Best complete or partial response (Objective response rate) | Yes | xx (xx%) |
| | No | xx (xx%) |
| | Missing value | xx - |

Table 61: Requirement for medical procedures (safety population- standard follow-up)

| | | V1 - End of<br>cycle 1<br>(N=xxx) | V2 - End of<br>cycle 2<br>(N=xxx) | V3 - End of<br>cycle 4<br>(N=xxx) | Standard follow-up<br>(N=xxx) |
|---|---|---|---|---|---|
| At least 1 consultation | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, at least 1 | Planned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| • | Unplanned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| At least 1 hospitalization | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| - | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If yes, at least 1 | Planned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| , . | Unplanned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| At least 1 hospitalization AND | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 consultation | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| At least 1 call to a health | Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| professional | No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

| | | V1 - End of<br>cycle 1<br>(N=xxx) | V2 - End of<br>cycle 2<br>(N=xxx) | V3 - End of<br>cycle 4<br>(N=xxx) | Standard follow-up<br>(N=xxx) |
|---|---|---|---|---|---|
| If yes, at least 1 | Planned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Unplanned | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Table 62: Patient adherence with treatment (safety population- standard follow-up)

| | | End of cycle 1<br>(N=xxx) | End of cycle 2<br>(N=xxx) | End of cycle<br>4<br>(N=xxx) |
|---|---|---|---|---|
| MMAS-4 score (adherence score)* | Number analyzed | xxx | xxx | xxx |
| | Mean (±SD) | xx (± xx) | xx (± xx) | xx (± xx) |
| | Median | XX | xx | XX |
| | Min-Max | xx - xx | xx - xx | xx - xx |
| Level of adherence | High: 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Mean: 1 or 2 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Low: 3 or 4 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Missing value | xx - | xx - | xx - |
| "Adherent" patient | Yes: 0 | xx (xx%) | xx (xx%) | xx (xx%) |
| - | No: >=1 | xx (xx%) | xx (xx%) | xx (xx%) |
| | Missing value | xx - | xx - | xx - |

### 10. REFERENCES

#### References – Adherence

- 1. Garber MC, Nau DP, Erickson SR, Aikens JE, Lawrence JB. The concordance of self-report with other measures of medication adherence: a summary of the literature. Medical care. 2004;42(7):649-52. Epub 2004/06/24.
- 2. Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Medical care. 1986;24(1):67-74. Epub 1986/01/01.
- 3. Landis JR, Koch GG. The Measurement of Observer Agreement for Categorical Data, Biometrics, 1977a, 33, 159-174.
- 4. Ravaud, A, et al. Real-life patterns of use and effectiveness of sunitinib in patients with metastatic renal cell carcinoma: The SANTORIN study. ASCO.
- 5. Natarajan N, Putnam RW, Yip AM. Family practice patients' adherence to statin medications. *Can Fam Physician*, 2007 December; 53(12): 2144–2145.
- 6. Tordoff JM, Bagge ML, Gray AR, Campbell AJ, Norris PT. Medicine-taking practices in community-dwelling people aged ≥ 75 years in New Zealand. *Age and Ageing*, 2010; 1–7.
- 7. Efficace F, Baccarani M, Rosti G, Castagnetti F, Breccia M et al. Investigating factors associated with adherence behavior in patients with chronic myeloid leukemia: an observational patient-centered outcome study. Br J Cancer., 2012 Sep 4;107(6):904-9
- 8. Noize P, Grelaud A, Bay JO, Chevreau C, Gross-Goupil M, Culine S et al. Real-life patterns of use, safety and effectiveness of sunitinib in first line therapy of metastatic renal cell carcinoma: the SANTORIN cohort study. pharmacoepidemiology and drug safety 2017; 26: 1561–1569.

### 11. Annexes

# 11.1. Interpretation of the Kappa coefficient

| Accord | Kappa |
|-----------|-------------|
| Excellent | ³ 0,81 |
| PPD | 0,80 - 0,61 |
| | 0,60 - 0,41 |
| 5954B | 0,40 - 0,21 |
| | 0,20 - 0,0 |
| | < 0,0 |

#### **Sources:**

Landis JR, Koch G.G. The Measurement of Observer Agreement for Categorical Data, *Biometrics*, 1977a, **33**, 159-174.

http://kappa.chez-alice.fr/Kappa\_2juges\_Def.htm

## 11.2. Definition of region indicators

Figure 4: Definition of region indicators

| Region (Insee 2016) | Département |
|---|---|
| PPD | 01, 03, 07, 15, 26, 38, 42, 43, 63, 69, 73, 74 |
| PPD | 21, 25, 39, 58, 70, 71, 89, 90 |
| PPD | 22, 29, 35, 56 |
| PPD | 18, 28, 36, 37, 41, 45 |
| PPD | 20 |
| PPD | 08, 10, 51, 52, 54, 55, 57, 67, 68, 88 |
| PPD | 02, 59, 60, 62, 80 |
| PPD | 91, 92, 75, 93, 77, 94, 95, 78 |
| PPD | 14, 27, 50, 61, 76 |
| PPD | 16, 17, 19, 23, 24, 33, 40, 47, 64, 79, 86, 87 |
| PPD | 09, 11, 12, 30, 31, 32, 34, 46, 48, 65, 66, 81, 82 |
| PPD | 44, 49, 53, 72, 85 |
| PPD | 04, 06, 13, 05, 83, 84, 980 (Monaco) |